CLINICAL TRIAL: NCT02509026
Title: A MULTICENTER OPEN-LABEL STUDY OF ETANERCEPT WITHDRAWAL AND RETREATMENT IN SUBJECTS WITH NON-RADIOGRAPHIC AXIAL SPONDYLOARTHRITIS WHO ACHIEVED ADEQUATE 24 WEEK RESPONSE
Brief Title: Etanercept Withdrawal And Retreament Study In Subjects With Nr-ax SpA
Acronym: RE-EMBARK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1801381; 2015-000541-24 (EudraCT Number)
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Spondylitis, Ankylosing
Keywords: non-radiographic axial spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Non-Radiographic Axial Spondyloarthritis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etanercept (Experimental): etanercept 50 mg QW
  Interventions: Biological: Etanercept

INTERVENTIONS:
Biological: Etanercept — 50 mg subcutaneous, once weekly, 24 weeks

SUMMARY:
The purpose of this study is to study the benefits and risks of etanercept withdrawal in patients who have achieved a significant clinical response.

DETAILED DESCRIPTION:
This multcenter, open-label, three period study will evaluate withdrawal and retreatment of etanercept in subjects with nr-ax SpA who achieved adequate response following 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of axial SpA duration of symptoms >3 months and <5 years back pain with a less than favorable response to NSAIDs

Exclusion Criteria:

* radiological sacroiliitis previous treatment with TNF inhibitor, biologic, immunosuppressive

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- United States (12):
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - Northwestern Medical Group; Division of Rheumatology, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Clinical and Translational Sciences Institute (NUCATS), Chicago, Illinois
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - Oregon Health and Science University Research Pharmacy, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Swedish Medical Center Investigational Drug Services Pharmacy, Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (9):
  - Genesis Research Services Pty Ltd, Broadmeadow, New South Wales
  - Hunter Imaging Group, Cardiff, New South Wales
  - Pacific Radiology, Maroochydore, Queensland
  - Rheumatology Research Centre, Maroochydore, Queensland
  - Benson Radiology, North Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - SKG Radiology Hollywood Hospital, Nedlands, Western Australia
  - SKG Radiology Subiaco, Subiaco, Western Australia
  - R.K. Will Pty Ltd, Victoria Park, Western Australia
- Belgium (2):
  - Private Practice Rheumatology, Sint-Niklaas, OVL
  - Reumaclinic, Genk
- Colombia (3):
  - Centro Integral de Reumatologia Reumalab S.A.S., Medellín, Antioquia
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Preventive Care SAS, Chía, Cundinamarca
- Czechia (5):
  - Revmatologicky ustav, Prague
  - Affidea Praha s.r.o., Prague
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
  - Uherskohradist' ska nemocnice a.s., Uherské Hradiště
  - Lekarna Hradebni s.r.o., Uherské Hradiště
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - HYKS, Meilahden kolmiosairaala, Helsinki
  - Kiljavan Laaketutkimus Oy, Hyvinkää
- France (8):
  - Service d'Imagerie Guilloz, Nancy
  - Hopital Cochin Pavillon Hardy B4, Paris
  - Pharmacie-Secteur Essais cliniques, Paris
  - CHU de Rennes, Hopital Sud, Rennes
  - CHU PURPAN, Hopital Pierre-Paul Riquet, Toulouse
  - Pharmacie, Toulouse
  - Pharmacie Essais cliniques, Vandœuvre-lès-Nancy
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Medizinische Klinik und Poliklinik IV, Munich, Bavaria
  - Rheumazentrum Ruhrgebiet, Herne, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin, Berlin
  - Apotheke am Tierpark, Berlin
  - Praxis für radiologische Diagnostik, Berlin
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Schlosspark-Klinik GmbH, Berlin
  - Mvz Agilomed, Chemnitz
  - Universitaetskliniken Koeln, Cologne
- Hungary (2):
  - Qualiclinic Kft., Budapest
  - VITAL MEDICAL CENTER Orvosi es Fogorvosi Kozpont, Veszprém
- Netherlands (2):
  - READE, Amsterdam
  - LUMC, Leiden
- Poland (14):
  - Nzoz McD Voxel, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela w Bydgoszczy, Klinika Reumatologii i Ukladowych Chorob, Bydgoszcz
  - Zaklad Radiologii i Diagnostyki Obrazowej, Bydgoszcz
  - Centrum Kliniczno-Badawcze J. Brzezicki, B. Gornikiewicz-Brzezicka Lekarze Spolka Partnerska, Elblag
  - Samodzielny Publiczny Zespol Opieki Zdrowotnej, Kościan
  - Reumed Sp z.o.o. Zespool Poradni Specjalistycznych Filia nr 1, Lublin
  - RCMed, Nowy Duninów
  - Diagnostic-Med Centrum Diagnostyki Radiologicznej, Poznan
  - RCMed, Sochaczew
  - SANUS Szpital Specjalistyczny Sp. z o.o., Stalowa Wola
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Medycyna Kliniczna, Warsaw
  - Reumatika-Centrum Reumatologii NZOZ, Warsaw
  - Centrum Medyczne OPOROW, Wroclaw
- Spain (5):
  - Complejo Hospitalario Universitario Santiago, Santiago de Compostela, A Coruna
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital San Rafael, A Coruña
  - Complejo Hospitalario Regional Virgen Macarena, Seville
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skanes University Hospital Malmo, Malmo
  - Akademiska sjukhuset, Uppsala
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Chung Shan Medical University, Taichung
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Van den Bosch F, Wei JC, Nash P, Blanco FJ, Graham D, Zang C, Arthur E, Borlenghi C, Tsekouras V, Vlahos B, Deodhar A. Etanercept Withdrawal and Retreatment in Nonradiographic Axial Spondyloarthritis: Results of RE-EMBARK, an Open-Label Phase IV Trial. J Rheumatol. 2023 Apr;50(4):478-487. doi: 10.3899/jrheum.220353. Epub 2022 Nov 15. PMID 36379575
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801381&StudyName=A%20Multicenter%20Open-label%20Study%20Of%20Etanercept%20Withdrawal%20And%20Retreatment%20In%20Subjects%20With%20Non-radiographic%20Axial%20Spondyloarthritis%20Who%20Achieved%20Adequate%2024%20Week%20Response

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first visit of the Period 3 (re-treatment period) might occur at the same time as a regularly scheduled visit during Period 2 (withdrawal period) or as an unscheduled visit for a participant who experienced flare during Period 2.
Groups:
- Etanercept: All enrolled participants with non-radiographic axial spondyloarthritis (nr-ax SpA) were treated for 24 weeks with 50-milligram (mg) weekly dose of Etanercept in Period 1 (Induction Period). Participants who achieved ankylosing spondylitis disease activity scale (ASDAS) C-reactive protein (CRP) level less than (<) 1.3 at Week 24 entered into Period 2 (Withdrawal Period). In this period, participants discontinued Etanercept for 40 weeks and participants who achieved an ASDAS erythrocyte sedimentation rate (ESR) level greater than or equal to (>=) 2.1 by Week 64, then entered into Period 3 (Retreatment Period) of 12 weeks, treated with 50 mg weekly doses, and then followed up until 28 days after last dose of Etanercept. Participants who did not qualify for Period 2 or 3 were followed up until 28 days after last dose of Etanercept.
Period: Induction Period (24 Weeks)
Arm/Group | Etanercept
Started | 210
Treated | 209
Completed | 188
Not Completed | 22
Not completed — Adverse Event | 5
Not completed — Eligibility Criteria | 5
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 1
Not completed — Other | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Enrolled but not treated | 1
Period: Withdrawal Period (40 Weeks)
Arm/Group | Etanercept
Started | 119 (Participants who completed Period 1 and achieved ASDAS-CRP<1.3 were eligible to enter into Period 2)
Completed | 112
Not Completed | 7
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 5
Period: Retreatment Period (12 Weeks)
Arm/Group | Etanercept
Started | 88 (Participants who completed Period 2 and achieved ASDAS-ESR>=2.1 were eligible to enter into Period 3)
Treated | 87
Completed | 84
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who took study drug and had 1 evaluation after baseline (Day 1).
Groups:
- Etanercept: All enrolled participants with nr-ax SpA were treated for 24 weeks with 50-mg weekly dose of Etanercept in Period 1 (Induction Period). Participants who achieved ASDAS CRP level < 1.3 at Week 24 entered into Period 2 (Withdrawal Period). In this period, participants discontinued Etanercept for 40 weeks and participants who achieved an ASDAS ESR level >= 2.1 by Week 64, then entered into Period 3 (Retreatment Period) of 12 weeks, treated with 50 mg weekly doses, and then followed up until 28 days after last dose of Etanercept. Participants who did not qualify for Period 2 or 3 were followed up until 28 days after last dose of Etanercept.
Arm/Group | Etanercept
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.1 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 112
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 186
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Flare Within 40 Weeks Following Withdrawal of 24 Weeks of Etanercept Treatment
Description: Participants who experienced ASDAS-Erythrocyte Sedimentation Rate (ESR) level of >=2.1 were defined as being flared. ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0 = no disease activity and 10= high disease activity. CRP measured in milligram per liter (mg/L) and ESR measured in millimeter per hour (mm/hr). Percentage of participants who flared within 40 weeks after the withdrawal of Etanercept treatment of 24 weeks in Induction period are reported in this outcome measure.
Time Frame: Within 40 weeks after Etanercept withdrawal (from Week 24 to Week 64)
Population: Full analysis set for period 2 included all participants who had at least one evaluation during period 2. Missing data was imputed using mixed last observation carried forward (LOCF).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants | 74.8 [66.30 to 82.04]

2. Secondary Outcome: Time to Flare Following Withdrawal of Etanercept Treatment
Description: Participants who experienced ASDAS-ESR level of >=2.1 were defined as being flared. Time to experience flare in participants was defined as time to achieve ASDAS-ESR level of >=2.1 after the withdrawal of Etanercept treatment of 24 weeks in induction period. ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0 = no disease activity and 10= high disease activity. CRP measured in mg/L and ESR measured in mm/hr.
Time Frame: Within 40 weeks after Etanercept withdrawal (from Week 24 to Week 64)
Population: Full analysis set for period 2 included all participants who had at least one evaluation during period 2.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 115
weeks | 16.1 [12.57 to 24.00]

3. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<)1.3: Observed Cases (OC): Period 1
Description: ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0= no disease activity and 10= high disease activity. CRP measured in mg/L and ESR measured in mm/hr. ASDAS ranged as inactive disease: 0 <= ASDAS-CRP <1.3; moderate disease activity: 1.3 <= ASDAS-CRP <2.1; high disease activity: 2.1 <= ASDAS-CRP <=3.5; very high disease activity: 3.5 < ASDAS-CRP.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Baseline: number analyzed (Participants) | 206
  Baseline | 0.5 [0.05 to 2.25]
  Week 4 | 14.4 [10.15 to 19.68]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 27.4 [21.55 to 33.82]
  Week 12: number analyzed (Participants) | 197
  Week 12 | 38.1 [31.50 to 44.99]
  Week 16: number analyzed (Participants) | 191
  Week 16 | 41.9 [35.05 to 48.96]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 62.6 [55.60 to 69.28]

4. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<)1.3: Observed Cases (OC): Period 2
Description: as for outcome 3
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: Full analysis set for Period 2 included all participants who had at least one evaluation during period 2. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 52.7 [43.43 to 61.89]
  Week 32: number analyzed (Participants) | 93
  Week 32 | 45.2 [35.32 to 55.29]
  Week 40: number analyzed (Participants) | 66
  Week 40 | 48.5 [36.71 to 60.39]
  Week 48: number analyzed (Participants) | 50
  Week 48 | 42.0 [29.09 to 55.81]
  Week 56: number analyzed (Participants) | 41
  Week 56 | 56.1 [40.93 to 70.44]
  Week 64: number analyzed (Participants) | 34
  Week 64 | 55.9 [39.28 to 71.53]

5. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<)1.3: Observed Cases (OC): Period 3
Description: as for outcome 3
Time Frame: Week 68, 72, 76
Population: Full analysis set for Period 3 included all participants who took study retreatment medication and had at least one evaluation after restarting active therapy. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 68: number analyzed (Participants) | 84
  Week 68 | 53.6 [42.94 to 63.96]
  Week 72: number analyzed (Participants) | 86
  Week 72 | 61.6 [51.10 to 71.38]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 62.4 [51.78 to 72.10]

6. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<) 1.3: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 3
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Missing data was imputed using mixed LOCF. Overall Number of Participants Analyzed" = participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Baseline: number analyzed (Participants) | 206
  Baseline | 0.5 [0.05 to 2.25]
  Week 4 | 14.4 [10.15 to 19.68]
  Week 8 | 27.4 [21.68 to 33.75]
  Week 12 | 36.5 [30.22 to 43.23]
  Week 16 | 40.4 [33.89 to 47.15]
  Week 24 | 58.7 [51.88 to 65.19]

7. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<) 1.3: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 3
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: Full analysis set for Period 2 included all participants who had at least one evaluation during period 2. Missing data was imputed using mixed LOCF. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 52.7 [43.43 to 61.89]
  Week 32: number analyzed (Participants) | 113
  Week 32 | 39.8 [31.15 to 49.01]
  Week 40: number analyzed (Participants) | 113
  Week 40 | 34.5 [26.23 to 43.58]
  Week 48: number analyzed (Participants) | 113
  Week 48 | 26.5 [19.07 to 35.21]
  Week 56: number analyzed (Participants) | 113
  Week 56 | 29.2 [21.42 to 38.03]
  Week 64: number analyzed (Participants) | 113
  Week 64 | 24.8 [17.52 to 33.31]

8. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Less Than (<) 1.3: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 3
Time Frame: Week 68, 72, 76
Population: Full analysis set for Period 3 included all participants who took study retreatment medication and had at least one evaluation after restarting active therapy. Missing data was imputed using mixed LOCF. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 68: number analyzed (Participants) | 85
  Week 68 | 52.9 [42.38 to 63.31]
  Week 72 | 60.9 [50.45 to 70.68]
  Week 76 | 62.1 [51.61 to 71.74]

9. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Observed Cases (OC): Period 1
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, total back pain, function (from [Bath Ankylosing Spondylitis Functional Index] BASFI) and inflammation (from [Bath Ankylosing Spondylitis Disease Activity Index] BASDAI). ASAS 20 responders were defined as participants with at least 20% improvement from baseline in disease activity and an absolute change of at least 1 unit on a 0 to 10 cm scale (0=no disease activity; 10=high disease activity, where higher scores indicated higher disease activity) in 3 or more domains, and no worsening of >=20% and absolute change 1 unit in the remaining domain. All 4 domains were measured on a 0-100 millimeter (mm) scale (0= no disease activity; 100 = high disease activity, where higher scores indicated higher disease activity). These scores were then converted to 0-10 cm scale for assessment of ASAS 20.
Time Frame: Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Here, "Overall Number of Participants Analyzed" signifies participants evaluable at this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 58.7 [51.88 to 65.19]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 68.7 [62.01 to 74.77]
  Week 12: number analyzed (Participants) | 198
  Week 12 | 71.7 [65.16 to 77.64]
  Week 16: number analyzed (Participants) | 192
  Week 16 | 78.1 [71.88 to 83.52]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 85.8 [80.30 to 90.20]

10. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Observed Cases (OC): Period 2
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, total back pain, function (from BASFI) and inflammation (from BASDAI). ASAS 20 responders were defined as participants with at least 20% improvement from baseline in disease activity and an absolute change of at least 1 unit on a 0 to 10 cm scale (0=no disease activity; 10=high disease activity, where higher scores indicated higher disease activity) in 3 or more domains, and no worsening of >=20% and absolute change 1 unit in the remaining domain. All 4 domains were measured on a 0-100 millimeter (mm) scale (0= no disease activity; 100 = high disease activity, where higher scores indicated higher disease activity). These scores were then converted to 0-10 cm scale for assessment of ASAS 20.
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 86.0 [78.21 to 91.74]
  Week 32: number analyzed (Participants) | 81
  Week 32 | 88.9 [80.71 to 94.36]
  Week 40: number analyzed (Participants) | 59
  Week 40 | 83.1 [72.02 to 90.94]
  Week 48: number analyzed (Participants) | 47
  Week 48 | 91.5 [81.02 to 97.06]
  Week 56: number analyzed (Participants) | 35
  Week 56 | 91.4 [78.86 to 97.53]
  Week 64: number analyzed (Participants) | 27
  Week 64 | 92.6 [78.30 to 98.43]

11. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Observed Cases (OC): Period 3
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, total back pain, function (from BASFI) and inflammation (from BASDAI). ASAS 20 responders: participants with at least 20% improvement from baseline in disease activity and an absolute change of at least 1 unit on 0 to 10 cm scale(0=no disease activity; 10=high disease activity, where higher scores indicated higher disease activity)in 3 or more domains, and no worsening of >=20% and absolute change 1 unit in the remaining domain. All 4 domains measured on 0-100 millimeter (mm) scale (0= no disease activity; 100 = high disease activity, where higher scores indicated higher disease activity). These scores were then converted to 0-10 cm scale for assessment of ASAS 20.
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 33.3 [14.03 to 58.42]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 80.0 [70.58 to 87.42]
  Week 72 | 81.6 [72.51 to 88.65]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 87.1 [78.72 to 92.93]

12. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 10
Time Frame: Week 4, 8, 12, 16, 24
Population: FAS for Period 1 included all participants who took study medication and had one evaluation after baseline. Missing data was imputed using mixed LOCF. "Overall Number of Participants Analyzed" included participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 58.7 [51.88 to 65.19]
  Week 8 | 68.8 [62.23 to 74.76]
  Week 12 | 71.2 [64.74 to 76.99]
  Week 16 | 76.4 [70.34 to 81.82]
  Week 24 | 83.2 [77.65 to 87.78]

13. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 10
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 86.0 [78.21 to 91.74]
  Week 32: number analyzed (Participants) | 102
  Week 32 | 84.3 [76.34 to 90.37]
  Week 40: number analyzed (Participants) | 102
  Week 40 | 79.4 [70.81 to 86.37]
  Week 48: number analyzed (Participants) | 102
  Week 48 | 79.4 [70.81 to 86.37]
  Week 56: number analyzed (Participants) | 102
  Week 56 | 78.4 [69.73 to 85.55]
  Week 64: number analyzed (Participants) | 102
  Week 64 | 77.5 [68.65 to 84.72]

14. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS 20) Response: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 11
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 33.3 [14.03 to 58.42]
  Week 68: number analyzed (Participants) | 86
  Week 68 | 79.1 [69.60 to 86.62]
  Week 72 | 81.6 [72.51 to 88.65]
  Week 76 | 86.2 [77.82 to 92.23]

15. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Last Observation Carried Forward (LOCF): Period 1
Description: ASAS measures symptomatic improvement in AS in 4 domains: participant global assessment of disease activity, total back pain, function (from BASFI) and inflammation (from BASDAI). ASAS 40 responders were defined as participants with at least 40% and absolute improvement of at least 2 units on a 0 to 10 cm scale (converted from 0 to 100 mm) or an improvement of 100% for those domains that have a baseline score <2 in at least 3 of the 4 domains: participant assessment of disease activity, mean of participants assessment of total back pain, function represented by the BASFI score, inflammation represented by the mean of the two morning stiffness-related BASDAI scores. No worsening at all in any of the domains. Each domain was measured on a 0-100 mm scale (0=no disease activity; 100 = high disease activity, where higher scores indicated higher disease activity). These scores were then converted to 0-10 cm scale for assessment of ASAS 40.
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 34.6 [28.40 to 41.26]
  Week 8 | 49.0 [42.30 to 55.81]
  Week 12 | 51.0 [44.19 to 57.70]
  Week 16 | 61.1 [54.32 to 67.49]
  Week 24 | 71.6 [65.24 to 77.43]

16. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 15
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 77.0 [68.06 to 84.40]
  Week 32: number analyzed (Participants) | 102
  Week 32 | 72.5 [63.35 to 80.49]
  Week 40: number analyzed (Participants) | 102
  Week 40 | 69.6 [60.23 to 77.89]
  Week 48: number analyzed (Participants) | 102
  Week 48 | 64.7 [55.12 to 73.47]
  Week 56: number analyzed (Participants) | 102
  Week 56 | 66.7 [57.15 to 75.25]
  Week 64: number analyzed (Participants) | 102
  Week 64 | 62.7 [53.11 to 71.67]

17. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 15
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 20.0 [5.98 to 44.36]
  Week 68: number analyzed (Participants) | 86
  Week 68 | 67.4 [57.09 to 76.64]
  Week 72 | 74.7 [64.88 to 82.94]
  Week 76 | 77.0 [67.38 to 84.88]

18. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Observed Cases (OC): Period 1
Description: as for outcome 15
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 34.6 [28.40 to 41.26]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 49.3 [42.39 to 56.13]
  Week 12: number analyzed (Participants) | 198
  Week 12 | 52.5 [45.58 to 59.40]
  Week 16: number analyzed (Participants) | 192
  Week 16 | 64.1 [57.11 to 70.60]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 75.8 [69.34 to 81.46]

19. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Observed Cases (OC): Period 2
Description: as for outcome 15
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 77.0 [68.06 to 84.40]
  Week 32: number analyzed (Participants) | 81
  Week 32 | 77.8 [67.85 to 85.76]
  Week 40: number analyzed (Participants) | 59
  Week 40 | 74.6 [62.48 to 84.33]
  Week 48: number analyzed (Participants) | 47
  Week 48 | 74.5 [60.81 to 85.22]
  Week 56: number analyzed (Participants) | 35
  Week 56 | 82.9 [68.03 to 92.51]
  Week 64: number analyzed (Participants) | 27
  Week 64 | 74.1 [55.71 to 87.58]

20. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society 40 (ASAS 40) Response: Observed Cases (OC): Period 3
Description: as for outcome 15
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 20.0 [5.98 to 44.36]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 68.2 [57.86 to 77.40]
  Week 72 | 74.7 [64.88 to 82.94]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 78.8 [69.27 to 86.46]

21. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Last Observation Carried Forward (LOCF): Period 1
Description: ASAS partial remission was defined as a score of 2 units or less (on a scale of 0-10 cm, where 0 = no disease activity and 10 = high disease activity) in each of the 4 domains of ASAS: participant global assessment of disease activity, total back pain, function (from BASFI) and inflammation (from BASDAI). Each domain was measured on a 0-100 mm scale (0=no disease activity; 100 = high disease activity, where higher scores indicated higher disease activity). Reported values were then converted into cm for analysis.
Time Frame: Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Missing data was imputed using mixed LOCF. Here, "Overall Number of Participants Analyzed" included participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 19.2 [14.32 to 24.99]
  Week 8 | 29.8 [23.90 to 36.27]
  Week 12 | 37.0 [30.67 to 43.72]
  Week 16 | 40.9 [34.35 to 47.63]
  Week 24 | 58.2 [51.39 to 64.73]

22. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 21
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 63.0 [53.28 to 71.98]
  Week 32: number analyzed (Participants) | 102
  Week 32 | 53.9 [44.25 to 63.37]
  Week 40: number analyzed (Participants) | 102
  Week 40 | 48.0 [38.51 to 57.68]
  Week 48: number analyzed (Participants) | 102
  Week 48 | 41.2 [31.98 to 50.86]
  Week 56: number analyzed (Participants) | 102
  Week 56 | 44.1 [34.76 to 53.81]
  Week 64: number analyzed (Participants) | 102
  Week 64 | 41.2 [31.98 to 50.86]

23. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 21
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 0.0 [0.00 to 15.18]
  Week 68: number analyzed (Participants) | 86
  Week 68 | 45.3 [35.13 to 55.88]
  Week 72 | 55.2 [44.70 to 65.31]
  Week 76 | 52.9 [42.43 to 63.13]

24. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Observed Cases (OC): Period 1
Description: as for outcome 21
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 19.2 [14.32 to 24.99]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 30.3 [24.31 to 36.95]
  Week 12: number analyzed (Participants) | 198
  Week 12 | 38.9 [32.30 to 45.80]
  Week 16: number analyzed (Participants) | 192
  Week 16 | 42.7 [35.86 to 49.77]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 62.1 [55.07 to 68.78]

25. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Observed Cases (OC): Period 2
Description: as for outcome 21
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 100
  Week 28 | 63.0 [53.28 to 71.98]
  Week 32: number analyzed (Participants) | 81
  Week 32 | 58.0 [47.15 to 68.34]
  Week 40: number analyzed (Participants) | 59
  Week 40 | 59.3 [46.59 to 71.16]
  Week 48: number analyzed (Participants) | 47
  Week 48 | 51.1 [37.07 to 64.93]
  Week 56: number analyzed (Participants) | 35
  Week 56 | 68.6 [52.20 to 82.02]
  Week 64: number analyzed (Participants) | 27
  Week 64 | 70.4 [51.75 to 84.88]

26. Secondary Outcome: Percentage of Participants Who Achieved Assessment of Spondyloarthritis Society (ASAS) Partial Remission: Observed Cases (OC): Period 3
Description: as for outcome 21
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 0.0 [0.00 to 15.18]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 45.9 [35.57 to 56.47]
  Week 72 | 55.2 [44.70 to 65.31]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 52.9 [42.38 to 63.31]

27. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-C-Reactive Protein (CRP) Score: Last Observation Carried Forward (LOCF): Period 1
Description: ASDAS: score combining assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on VAS ranging 0-10 cm, where 0= no disease activity and 10= high disease activity. CRP measured in mg/L and ESR measured in mm/hr. ASDAS ranged as inactive disease: 0<= ASDAS-CRP <1.3; moderate disease activity: 1.3<= ASDAS-CRP <2.1; high disease activity: 2.1<= ASDAS-CRP <=3.5; very high disease activity: 3.5< ASDAS-CRP. The ASDAS-CRP is calculated with the following equation: 0.121*total back pain+0.110*participant global+0.073*peripheral pain/swelling+0.058*duration of morning stiffness+0.579*Ln(CRP+1), Ln represents the natural logarithm.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Missing data was imputed using mixed LOCF. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 3.54 (0.87)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -1.27 (1.02)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -1.53 (1.09)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -1.62 (1.15)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -1.77 (1.13)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -2.02 (1.15)

28. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-C-Reactive Protein (CRP) Score: Last Observation Carried Forward (LOCF): Period 2
Description: ASDAS: score combining assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on VAS ranging 0-10 cm,where 0= no disease activity and 10= high disease activity.CRP measured in mg/L and ESR measured in mm/hr. ASDAS ranged as inactive disease: 0<= ASDAS-CRP <1.3; moderate disease activity: 1.3<= ASDAS-CRP <2.1; high disease activity: 2.1<= ASDAS-CRP <=3.5; very high disease activity: 3.5< ASDAS-CRP. The ASDAS-CRP is calculated with the following equation: 0.121*total back pain+0.110*participant global+0.073*peripheral pain/swelling+0.058*duration of morning stiffness+0.579*Ln(CRP+1), Ln represents the natural logarithm.
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.90 (0.20)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 1 Baseline | -1.83 (1.14)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 2 Baseline | 0.66 (0.89)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 113
  Change at Week 32 from Period 1 Baseline | -1.54 (1.17)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 32 from Period 2 Baseline | 0.96 (1.03)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 113
  Change at Week 40 from Period 1 Baseline | -1.36 (1.18)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 40 from Period 2 Baseline | 1.14 (1.07)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 113
  Change at Week 48 from Period 1 Baseline | -1.22 (1.18)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 48 from Period 2 Baseline | 1.29 (1.06)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 113
  Change at Week 56 from Period 1 Baseline | -1.17 (1.18)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 56 from Period 2 Baseline | 1.34 (1.07)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 113
  Change at Week 64 from Period 1 Baseline | -1.05 (1.16)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 64 from Period 2 Baseline | 1.46 (1.07)

29. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Score: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 27
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Period 3: Baseline (last visit before retreatment), Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 2.97 (0.91)
  Change at Week 64 from Period 1 baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 baseline | -0.44 (1.45)
  Change at Week 64 from Period 2 baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 baseline | 2.08 (0.80)
  Change at Week 64 from Period 3 baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 baseline | 0.23 (0.68)
  Change at Week 68 from Period 1 baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 baseline | -1.92 (1.06)
  Change at Week 68 from Period 2 baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 baseline | 0.67 (0.72)
  Change at Week 68 from Period 3 baseline: number analyzed (Participants) | 83
  Change at Week 68 from Period 3 baseline | -1.41 (0.98)
  Change at Week 72 from Period 1 baseline | -2.09 (1.02)
  Change at Week 72 from Period 2 baseline | 0.50 (0.69)
  Change at Week 72 from Period 3 baseline: number analyzed (Participants) | 85
  Change at Week 72 from Period 3 baseline | -1.58 (0.99)
  Change at Week 76 from Period 1 baseline | -2.12 (1.06)
  Change at Week 76 from Period 2 baseline | 0.47 (0.68)
  Change at Week 76 from Period 3 baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 3 baseline | -1.61 (1.04)

30. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Score: Observed Cases (OC): Period 1
Description: as for outcome 27
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: Full analysis set for Period 1 included all participants who took study medication and had one evaluation after baseline. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 3.54 (0.87)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -1.27 (1.02)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -1.54 (1.10)
  Change at week 12: number analyzed (Participants) | 197
  Change at week 12 | -1.66 (1.15)
  Change at week 16: number analyzed (Participants) | 191
  Change at week 16 | -1.85 (1.12)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -2.13 (1.09)

31. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Score: Observed Cases (OC): Period 2
Description: as for outcome 27
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.90 (0.20)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 1 Baseline | -1.83 (1.14)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 2 Baseline | 0.66 (0.89)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -1.76 (1.09)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 0.77 (0.93)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 66
  Change at Week 40 from Period 1 Baseline | -1.65 (1.09)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 40 from Period 2 Baseline | 0.74 (0.90)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 50
  Change at Week 48 from Period 1 Baseline | -1.59 (1.05)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 50
  Change at Week 48 from Period 2 Baseline | 0.78 (0.91)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 1 Baseline | -1.68 (1.04)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 2 Baseline | 0.63 (0.83)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -1.46 (1.08)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 0.74 (1.02)

32. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Score: Observed Cases (OC): Period 3
Description: as for outcome 27
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Period 3 Baseline (last visit before retreatment), Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 2.97 (0.91)
  Change at Week 64 from Period 1 baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 baseline | -0.44 (1.45)
  Change at Week 64 from Period 2 baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 baseline | 2.08 (0.80)
  Change at Week 64 from Period 3 baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 baseline | 0.23 (0.68)
  Change at Week 68 from Period 1 baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 1 baseline | -1.94 (1.05)
  Change at Week 68 from Period 2 baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 2 baseline | 0.65 (0.69)
  Change at Week 68 from Period 3 baseline: number analyzed (Participants) | 82
  Change at Week 68 from Period 3 baseline | -1.43 (0.97)
  Change at Week 72 from Period 1 baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 1 baseline | -2.11 (1.00)
  Change at Week 72 from Period 2 baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 2 baseline | 0.47 (0.65)
  Change at Week 72 from Period 3 baseline: number analyzed (Participants) | 84
  Change at Week 72 from Period 3 baseline | -1.61 (0.97)
  Change at Week 76 from Period 1 baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 baseline | -2.17 (1.03)
  Change at Week 76 from Period 2 baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 baseline | 0.45 (0.64)
  Change at Week 76 from Period 3 baseline: number analyzed (Participants) | 83
  Change at Week 76 from Period 3 baseline | -1.65 (1.02)

33. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) Erythrocyte Sedimentation Rate (ESR) Score: Last Observation Carried Forward (LOCF): Period 1
Description: ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0 = no disease activity and 100= high disease activity. CRP measured in mg/L and ESR measured in mm/hr. ASDAS-ESR was calculated with the following equation: 0.8*total back pain+0.11*participant global+0.09*peripheral pain/swelling+0.07*duration of morning stiffness+ 0.29*ESR^1/2. ASDAS ranged as inactive disease: 0 <= ASDAS-ESR <1.3; active disease: 1.3 <= ASDAS-ESR =<2.1.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 3.59 (0.90)
  Change at week 4: number analyzed (Participants) | 204
  Change at week 4 | -1.27 (0.98)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -1.56 (1.08)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -1.70 (1.15)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -1.81 (1.12)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -2.05 (1.17)

34. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-Erythrocyte Sedimentation Rate (ESR) Score: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 33
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.92 (0.37)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -1.81 (1.17)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 0.68 (0.90)
  Change at Week 32 from Period 1 Baseline | -1.58 (1.22)
  Change at Week 32 from Period 2 Baseline | 0.93 (1.03)
  Change at Week 40 from Period 1 Baseline | -1.34 (1.23)
  Change at Week 40 from Period 2 Baseline | 1.17 (1.05)
  Change at Week 48 from Period 1 Baseline | -1.16 (1.22)
  Change at Week 48 from Period 2 Baseline | 1.34 (1.05)
  Change at Week 56 from Period 1 Baseline | -1.11 (1.22)
  Change at Week 56 from Period 2 Baseline | 1.40 (1.07)
  Change at Week 64 from Period 1 Baseline | -0.98 (1.21)
  Change at Week 64 from Period 2 Baseline | 1.52 (1.12)

35. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-Erythrocyte Sedimentation Rate (ESR) Score: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 33
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline | 3.15 (0.72)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -0.54 (1.50)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 2 Baseline | 2.05 (0.84)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 0.10 (0.71)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -1.97 (1.01)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 0.65 (0.77)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 3 Baseline | -1.60 (0.85)
  Change at Week 72 from Period 1 Baseline | -2.15 (1.05)
  Change at Week 72 from Period 2 Baseline | 0.46 (0.74)
  Change at Week 72 from Period 3 Baseline | -1.77 (0.87)
  Change at Week 76 from Period 1 Baseline | -2.21 (1.09)
  Change at Week 76 from Period 2 Baseline | 0.41 (0.64)
  Change at Week 76 from Period 3 Baseline | -1.83 (0.90)

36. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) Erythrocyte Sedimentation Rate (ESR) Score: Observed Cases (OC): Period 1
Description: as for outcome 33
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 3.59 (0.90)
  Change at week 4: number analyzed (Participants) | 204
  Change at week 4 | -1.27 (0.98)
  Change at week 8: number analyzed (Participants) | 200
  Change at week 8 | -1.57 (1.09)
  Change at week 12: number analyzed (Participants) | 195
  Change at week 12 | -1.75 (1.16)
  Change at week 16: number analyzed (Participants) | 190
  Change at week 16 | -1.89 (1.11)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -2.16 (1.12)

37. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-Erythrocyte Sedimentation Rate (ESR) Score: Observed Cases (OC): Period 2
Description: as for outcome 33
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.92 (0.37)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -1.81 (1.17)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 0.68 (0.90)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 1 Baseline | -1.81 (1.12)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 2 Baseline | 0.70 (0.90)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 1 Baseline | -1.59 (1.13)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 2 Baseline | 0.77 (0.91)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -1.58 (1.11)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 0.81 (1.01)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 1 Baseline | -1.71 (1.04)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 2 Baseline | 0.56 (0.83)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -1.52 (1.16)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 0.73 (1.23)

38. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)-Erythrocyte Sedimentation Rate (ESR) Score: Observed Cases (OC): Period 3
Description: as for outcome 33
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline | 3.15 (0.72)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -0.54 (1.50)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 2 Baseline | 2.05 (0.84)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 0.10 (0.71)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -1.99 (1.01)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 0.63 (0.74)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 3 Baseline | -1.62 (0.83)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 1 Baseline | -2.17 (1.04)
  Change at Week 72 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 2 Baseline | 0.43 (0.69)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -1.80 (0.84)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 1 Baseline | -2.22 (1.07)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 2 Baseline | 0.39 (0.59)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 3 Baseline | -1.85 (0.88)

39. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Last Observation Carried Forward (LOCF): Period 1
Description: Major improvement in ASDAS-CRP was defined as decrease from baseline >= 2.0 units. ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0= no disease activity and 10= high disease activity. CRP measured in mg/L and ESR measured in mm/hr. The ASDAS-CRP is calculated with the following equation: 0.121*total back pain+0.110*participant global+0.073*peripheral pain/swelling+0.058*duration of morning stiffness+0.579*Ln(CRP+1), Ln represents the natural logarithm.
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 26.0 [20.36 to 32.22]
  Week 8 | 32.2 [26.14 to 38.77]
  Week 12 | 36.1 [29.76 to 42.74]
  Week 16 | 39.9 [33.43 to 46.66]
  Week 24 | 49.0 [42.30 to 55.81]

40. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 39
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 43.6 [34.63 to 52.97]
  Week 32: number analyzed (Participants) | 113
  Week 32 | 34.5 [26.23 to 43.58]
  Week 40: number analyzed (Participants) | 113
  Week 40 | 30.1 [22.22 to 38.97]
  Week 48: number analyzed (Participants) | 113
  Week 48 | 25.7 [18.30 to 34.26]
  Week 56: number analyzed (Participants) | 113
  Week 56 | 22.1 [15.24 to 30.42]
  Week 64: number analyzed (Participants) | 113
  Week 64 | 18.6 [12.25 to 26.50]

41. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 39
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 6.7 [0.73 to 27.18]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 41.2 [31.15 to 51.79]
  Week 72 | 55.2 [44.70 to 65.31]
  Week 76 | 54.0 [43.56 to 64.22]

42. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Observed Cases (OC): Period 1
Description: as for outcome 39
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 26.0 [20.36 to 32.22]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 32.8 [26.62 to 39.54]
  Week 12: number analyzed (Participants) | 197
  Week 12 | 38.1 [31.50 to 44.99]
  Week 16: number analyzed (Participants) | 191
  Week 16 | 42.4 [35.56 to 49.49]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 52.6 [45.54 to 59.65]

43. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Observed Cases (OC): Period 2
Description: as for outcome 39
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 43.6 [34.63 to 52.97]
  Week 32: number analyzed (Participants) | 93
  Week 32 | 39.8 [30.27 to 49.92]
  Week 40: number analyzed (Participants) | 66
  Week 40 | 37.9 [26.90 to 49.90]
  Week 48: number analyzed (Participants) | 50
  Week 48 | 34.0 [22.06 to 47.74]
  Week 56: number analyzed (Participants) | 41
  Week 56 | 31.7 [19.08 to 46.82]
  Week 64: number analyzed (Participants) | 34
  Week 64 | 23.5 [11.80 to 39.55]

44. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Major Improvement: Observed Cases (OC): Period 3
Description: as for outcome 39
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 6.7 [0.73 to 27.18]
  Week 68: number analyzed (Participants) | 84
  Week 68 | 41.7 [31.55 to 52.34]
  Week 72: number analyzed (Participants) | 86
  Week 72 | 55.8 [45.27 to 65.97]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 55.3 [44.70 to 65.54]

45. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Last Observation Carried Forward (LOCF): Period 1
Description: ASDAS-CRP clinically important improvement was defined as a decrease from baseline of >=1.1 units. ASDAS is a score combining the assessment of back pain, peripheral pain/swelling, duration of morning stiffness, participant global assessment of disease activity and CRP or ESR. All parameters other than CRP or ESR assessed on a VAS ranging from 0-10 cm, where 0= no disease activity and 10= high disease activity. CRP measured in mg/L and ESR measured in mm/hr. The ASDAS-CRP is calculated with the following equation: 0.121*total back pain+0.110* participant global+0.073*peripheral pain/swelling+0.058*duration of morning stiffness+0.579*Ln (CRP+1), Ln represents the natural logarithm.
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 55.8 [48.98 to 62.40]
  Week 8 | 64.4 [57.75 to 70.69]
  Week 12 | 63.9 [57.26 to 70.24]
  Week 16 | 71.6 [65.24 to 77.43]
  Week 24 | 77.4 [71.37 to 82.68]

46. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 45
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 74.5 [65.84 to 81.98]
  Week 32: number analyzed (Participants) | 113
  Week 32 | 70.8 [61.97 to 78.58]
  Week 40: number analyzed (Participants) | 113
  Week 40 | 59.3 [50.09 to 68.02]
  Week 48: number analyzed (Participants) | 113
  Week 48 | 55.8 [46.55 to 64.67]
  Week 56: number analyzed (Participants) | 113
  Week 56 | 54.9 [45.67 to 63.82]
  Week 64: number analyzed (Participants) | 113
  Week 64 | 50.4 [41.31 to 59.55]

47. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 45
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 26.7 [9.74 to 51.66]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 80.0 [70.58 to 87.42]
  Week 72 | 82.8 [73.82 to 89.56]
  Week 76 | 79.3 [69.93 to 86.78]

48. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Observed Cases (OC): Period 1
Description: as for outcome 45
Time Frame: Week 4, 8, 12, 16, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 55.8 [48.98 to 62.40]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 64.7 [57.90 to 71.04]
  Week 12: number analyzed (Participants) | 197
  Week 12 | 65.5 [58.66 to 71.86]
  Week 16: number analyzed (Participants) | 191
  Week 16 | 74.3 [67.82 to 80.14]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 81.1 [75.04 to 86.13]

49. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Observed Cases (OC): Period 2
Description: as for outcome 45
Time Frame: Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 110
  Week 28 | 74.5 [65.84 to 81.98]
  Week 32: number analyzed (Participants) | 93
  Week 32 | 79.6 [70.55 to 86.79]
  Week 40: number analyzed (Participants) | 66
  Week 40 | 68.2 [56.35 to 78.46]
  Week 48: number analyzed (Participants) | 50
  Week 48 | 72.0 [58.58 to 82.96]
  Week 56: number analyzed (Participants) | 41
  Week 56 | 78.0 [63.75 to 88.55]
  Week 64: number analyzed (Participants) | 34
  Week 64 | 70.6 [54.07 to 83.77]

50. Secondary Outcome: Percentage of Participants Who Achieved Ankylosing Spondylitis Disease Activity Score (ASDAS) C-Reactive Protein (CRP) Clinically Important Improvement: Observed Cases (OC): Period 3
Description: as for outcome 45
Time Frame: Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 26.7 [9.74 to 51.66]
  Week 68: number analyzed (Participants) | 84
  Week 68 | 81.0 [71.59 to 88.23]
  Week 72: number analyzed (Participants) | 86
  Week 72 | 83.7 [74.87 to 90.35]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 81.2 [71.90 to 88.37]

51. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Last Observation Carried Forward (LOCF): Period 1
Description: Participants assessed their nocturnal back pain over the last 48 hours on a 100 mm VAS scale ranged from 0 mm (none) to 100 mm (severe), where higher scores indicated more pain. The reported values were converted to centimeter (cm) for analysis.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 5.92 (2.52)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.53 (2.55)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -3.10 (2.76)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -3.25 (2.76)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -3.55 (2.67)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -4.14 (2.88)

52. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Last Observation Carried Forward (LOCF): Period 2
Description: Participants assessed their nocturnal back pain over the last 48 hours on a 100 mm VAS scale ranged from 0 mm (none) to 100 mm (severe), where higher scores indicated more pain. The reported values were converted to cm for analysis.
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.63 (1.07)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.77 (3.20)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 1.08 (2.33)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 1 Baseline | -3.05 (3.07)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 2 Baseline | 1.80 (2.65)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 1 Baseline | -2.64 (3.13)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 2 Baseline | 2.22 (2.89)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 1 Baseline | -2.32 (3.26)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 2 Baseline | 2.53 (2.93)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 1 Baseline | -2.11 (3.14)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 2 Baseline | 2.74 (3.00)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 1 Baseline | -1.77 (3.14)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 2 Baseline | 3.08 (3.06)

53. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 52
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 5.54 (2.63)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.28 (4.01)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.35 (2.87)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 1.29 (3.36)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -4.03 (2.81)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.33 (1.92)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 3 Baseline | -3.59 (2.64)
  Change at Week 72 from Period 1 Baseline | -4.43 (2.70)
  Change at Week 72 from Period 2 Baseline | 0.94 (1.87)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -3.96 (2.64)
  Change at Week 76 from Period 1 Baseline | -4.72 (2.82)
  Change at Week 76 from Period 2 Baseline | 0.64 (1.51)
  Change at Week 76 from Period 3 Baseline | -4.25 (2.74)

54. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Observed Cases (OC): Period 1
Description: as for outcome 52
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 5.92 (2.52)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.53 (2.55)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -3.10 (2.79)
  Change at week 12: number analyzed (Participants) | 198
  Change at week 12 | -3.32 (2.78)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -3.68 (2.68)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -4.32 (2.87)

55. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Observed Cases (OC): Period 2
Description: as for outcome 52
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.63 (1.07)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.77 (3.20)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 1.08 (2.33)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -3.50 (2.61)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 1.33 (2.38)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 1 Baseline | -3.12 (2.79)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 2 Baseline | 1.46 (2.67)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -3.03 (3.02)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 1.52 (2.73)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -3.22 (2.53)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 1.24 (2.69)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -2.28 (2.77)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.53 (3.01)

56. Secondary Outcome: Change From Baseline in Nocturnal Back Pain: Observed Cases (OC): Period 3
Description: as for outcome 52
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 5.54 (2.63)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.28 (4.01)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.35 (2.87)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 1.29 (3.36)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -4.07 (2.81)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.34 (1.93)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 3 Baseline | -3.62 (2.64)
  Change at Week 72 from Period 1 Baseline | -4.43 (2.70)
  Change at Week 72 from Period 2 Baseline | 0.94 (1.87)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -3.96 (2.64)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -4.84 (2.75)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 0.64 (1.51)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 3 Baseline | -4.36 (2.68)

57. Secondary Outcome: Change From Baseline in Total Back Pain: Last Observation Carried Forward (LOCF): Period 1
Description: Participants assessed their total back pain over the last 48 hours on a 100 mm VAS scale ranged from 0 mm (none) to 100 mm (severe), where higher scores indicated more pain. The reported values were converted to cm for analysis.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 5.98 (2.41)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.39 (2.36)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -2.96 (2.54)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -3.15 (2.60)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -3.44 (2.54)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -4.05 (2.79)

58. Secondary Outcome: Change From Baseline in Total Back Pain: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 57
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.71 (1.09)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.68 (3.04)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 1.09 (2.20)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 1 Baseline | -2.92 (3.06)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 2 Baseline | 1.84 (2.58)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 1 Baseline | -2.48 (3.17)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 2 Baseline | 2.28 (2.87)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 1 Baseline | -2.12 (3.19)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 2 Baseline | 2.64 (2.90)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 1 Baseline | -1.95 (3.16)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 2 Baseline | 2.81 (2.96)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 1 Baseline | -1.66 (3.13)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 2 Baseline | 3.10 (3.02)

59. Secondary Outcome: Change From Baseline in Total Back Pain: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 57
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 5.66 (2.55)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.10 (4.08)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.34 (2.70)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 1.07 (2.88)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -3.73 (2.66)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.35 (1.96)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 3 Baseline | -3.60 (2.55)
  Change at Week 72 from Period 1 Baseline | -4.21 (2.42)
  Change at Week 72 from Period 2 Baseline | 0.89 (1.81)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -4.03 (2.50)
  Change at Week 76 from Period 1 Baseline | -4.32 (2.70)
  Change at Week 76 from Period 2 Baseline | 0.77 (1.52)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 76 from Period 3 Baseline | -4.15 (2.72)

60. Secondary Outcome: Change From Baseline in Total Back Pain: Observed Cases (OC): Period 1
Description: as for outcome 57
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 5.98 (2.41)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.39 (2.36)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -2.97 (2.56)
  Change at week 12: number analyzed (Participants) | 198
  Change at week 12 | -3.23 (2.62)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -3.56 (2.53)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -4.24 (2.75)

61. Secondary Outcome: Change From Baseline in Total Back Pain: Observed Cases (OC): Period 2
Description: as for outcome 57
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.71 (1.09)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.68 (3.04)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 1.09 (2.20)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -3.43 (2.67)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 1.38 (2.35)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 1 Baseline | -2.97 (2.81)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 2 Baseline | 1.52 (2.69)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -2.91 (2.78)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 1.54 (2.65)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -3.15 (2.53)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 1.15 (2.52)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -2.56 (2.73)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.39 (2.96)

62. Secondary Outcome: Change From Baseline in Total Back Pain: Observed Cases (OC): Period 3
Description: as for outcome 57
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 5.66 (2.55)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.10 (4.08)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.34 (2.70)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 1.07 (2.88)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -3.76 (2.67)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.35 (1.97)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 3 Baseline | -3.63 (2.54)
  Change at Week 72 from Period 1 Baseline | -4.21 (2.42)
  Change at Week 72 from Period 2 Baseline | 0.89 (1.81)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -4.03 (2.50)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -4.41 (2.67)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 0.78 (1.53)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 3 Baseline | -4.24 (2.69)

63. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Observed Cases (OC): Period 1
Description: BASFI is composed of 10 questions related to the participant's ability to function. Each question scored by the participant on a 100 mm scale ranging from 0 (easy) to 100 (impossible), where higher scores indicated more difficulty in participant's ability to function. The BASFI total score calculated as mean of the scores for these 10 questions and converted to cm for analysis. BASFI total score was ranged from 0 (easy) to 10 (impossible), where higher scores indicated more difficulty in participant's ability to function due to ankylosing spondylitis.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 4.66 (2.21)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -1.62 (1.88)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -2.22 (2.21)
  Change at week 12: number analyzed (Participants) | 198
  Change at week 12 | -2.44 (2.34)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -2.73 (2.27)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -3.24 (2.57)

64. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Observed Cases (OC): Period 2
Description: as for outcome 63
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.59 (0.88)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.00 (2.78)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 0.90 (1.97)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -3.10 (2.52)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 0.88 (1.86)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 1 Baseline | -2.88 (2.41)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 68
  Change at Week 40 from Period 2 Baseline | 0.98 (1.63)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -2.84 (2.37)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 0.98 (1.76)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 1 Baseline | -2.97 (2.14)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 56 from Period 2 Baseline | 0.73 (1.57)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -2.33 (2.08)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.21 (2.41)

65. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Observed Cases (OC): Period 3
Description: as for outcome 63
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 4.14 (2.44)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.62 (3.52)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 3.11 (2.16)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 0.78 (2.73)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -2.99 (2.30)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.13 (1.58)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 3 Baseline | -2.41 (2.00)
  Change at Week 72 from Period 1 Baseline | -3.25 (2.35)
  Change at Week 72 from Period 2 Baseline | 0.84 (1.40)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -2.67 (2.22)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -3.47 (2.49)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 0.67 (1.30)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 76 from Period 3 Baseline | -2.89 (2.23)

66. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 63
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 4.66 (2.21)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -1.62 (1.88)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -2.23 (2.19)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -2.39 (2.31)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -2.65 (2.24)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -3.10 (2.54)

67. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 63
Time Frame: as for outcome 28
Population: Full analysis set for Period 2 included all participants who had at least one evaluation during period 2.Missing data was imputed using mixed LOCF. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.59 (0.88)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -3.00 (2.78)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 0.90 (1.97)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 1 Baseline | -2.54 (2.88)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 2 Baseline | 1.35 (2.22)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 1 Baseline | -2.21 (2.90)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 2 Baseline | 1.67 (2.29)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 1 Baseline | -1.97 (2.89)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 2 Baseline | 1.92 (2.36)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 1 Baseline | -1.85 (2.88)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 2 Baseline | 2.03 (2.40)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 1 Baseline | -1.62 (2.84)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 2 Baseline | 2.27 (2.51)

68. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI): Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 63
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 4.14 (2.44)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.62 (3.52)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 3.11 (2.16)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 0.78 (2.73)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -2.98 (2.29)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.14 (1.57)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 3 Baseline | -2.38 (2.01)
  Change at Week 72 from Period 1 Baseline | -3.25 (2.35)
  Change at Week 72 from Period 2 Baseline | 0.84 (1.40)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -2.67 (2.22)
  Change at Week 76 from Period 1 Baseline | -3.41 (2.49)
  Change at Week 76 from Period 2 Baseline | 0.68 (1.29)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 76 from Period 3 Baseline | -2.83 (2.24)

69. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score: Observed Cases (OC): Period 1
Description: BASDAI consisted of 6 questions related to disease activity. Each of the first 5 questions was scored by the participant on a 100 mm scale ranging from 0 (none) to 100 (very severe), where higher scores indicated more severe disease activity. The sixth question, related to duration of morning stiffness measured on a scale for 0 (0 hours) to 100 (2 hours), where higher scores indicated larger duration of morning stiffness. The BASDAI score was obtained by computing the mean score for the 2 questions related to morning stiffness (questions 5 [severity of morning stiffness] and 6 [duration of morning stiffness]) and then adding that value to the sum of the scores for the first 4 questions and then dividing the total by 5. This can be written as BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5. The BASDAI total score ranged from 0 to 10, where higher scores indicated more severe disease activity. The reported values were converted to cm for analysis.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 6.41 (1.80)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.39 (1.93)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -3.08 (2.17)
  Change at week 12: number analyzed (Participants) | 198
  Change at week 12 | -3.40 (2.37)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -3.91 (2.31)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -4.65 (2.36)

70. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score: Observed Cases (OC): Period 2
Description: as for outcome 69
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.63 (0.66)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -4.10 (2.61)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 1.38 (2.27)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 1 Baseline | -4.11 (2.40)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 2 Baseline | 1.37 (2.17)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 1 Baseline | -3.77 (2.46)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 2 Baseline | 1.60 (2.35)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -3.78 (2.32)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 1.65 (2.39)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -3.97 (2.18)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 1.20 (1.83)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -3.49 (2.47)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.49 (2.66)

71. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score: Observed Cases (OC): Period 3
Description: as for outcome 69
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline | 5.53 (2.24)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.92 (2.82)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.63 (2.14)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 0.37 (1.23)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -4.04 (2.10)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.66 (1.87)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 3 Baseline | -3.26 (2.15)
  Change at Week 72 from Period 1 Baseline | -4.47 (2.11)
  Change at Week 72 from Period 2 Baseline | 1.22 (1.73)
  Change at Week 72 from Period 3 Baseline | -3.65 (2.33)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -4.87 (2.21)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 0.91 (1.51)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 3 Baseline | -4.03 (2.38)

72. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 69
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 6.41 (1.80)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.39 (1.93)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -3.07 (2.16)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -3.34 (2.36)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -3.74 (2.36)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -4.41 (2.49)

73. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score:Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 69
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.63 (0.66)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -4.10 (2.61)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 1.38 (2.27)
  Change at Week 32 from Period 1 Baseline | -3.49 (2.75)
  Change at Week 32 from Period 2 Baseline | 1.99 (2.57)
  Change at Week 40 from Period 1 Baseline | -2.96 (2.80)
  Change at Week 40 from Period 2 Baseline | 2.52 (2.76)
  Change at Week 48 from Period 1 Baseline | -2.60 (2.76)
  Change at Week 48 from Period 2 Baseline | 2.88 (2.77)
  Change at Week 56 from Period 1 Baseline | -2.42 (2.75)
  Change at Week 56 from Period 2 Baseline | 3.06 (2.76)
  Change at Week 64 from Period 1 Baseline | -2.15 (2.71)
  Change at Week 64 from Period 2 Baseline | 3.33 (2.82)

74. Secondary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 69
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 87
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 86
  Period 3 Baseline | 5.53 (2.24)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.92 (2.82)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.63 (2.14)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 0.37 (1.23)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -4.01 (2.11)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.68 (1.86)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 3 Baseline | -3.20 (2.19)
  Change at Week 72 from Period 1 Baseline | -4.47 (2.11)
  Change at Week 72 from Period 2 Baseline | 1.22 (1.73)
  Change at Week 72 from Period 3 Baseline | -3.65 (2.33)
  Change at Week 76 from Period 1 Baseline | -4.78 (2.26)
  Change at Week 76 from Period 2 Baseline | 0.91 (1.51)
  Change at Week 76 from Period 3 Baseline | -3.96 (2.42)

75. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): Observed Cases (OC): Period 1
Description: 50% improvement from baseline in BASDAI: percentage of participants who achieved 50% decrease from baseline in their BASDAI total score. BASDAI consisted: 6 questions (Q) related to disease activity. Each of first 5 questions was scored by participant on 100 mm scale, range 0=none to 100=very severe, higher scores = more severe disease activity. Sixth question: duration of morning stiffness, was on scale for 0=0 hours to 100=2 hours, higher scores = larger duration of morning stiffness. BASDAI score was obtained by computing mean score for 2 questions related to morning stiffness (Q5 [severity of morning stiffness], Q6 [duration of morning stiffness]) and adding that value to sum of the scores for first 4Q and then dividing total by 5. BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5. BASDAI total score ranged from 0 to 10, higher scores = more severe disease activity. Reported values were converted to cm for analysis. Improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 33.7 [27.49 to 40.27]
  Week 8: number analyzed (Participants) | 201
  Week 8 | 50.7 [43.87 to 57.61]
  Week 12: number analyzed (Participants) | 198
  Week 12 | 57.1 [50.12 to 63.82]
  Week 16: number analyzed (Participants) | 192
  Week 16 | 66.7 [59.79 to 73.05]
  Week 24: number analyzed (Participants) | 190
  Week 24 | 78.9 [72.74 to 84.28]

76. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): Observed Cases (OC): Period 2
Description: 50% improvement from baseline in BASDAI: percentage of participants who achieved 50% decrease from baseline in their BASDAI total score. BASDAI consisted: 6 questions (Q) related to disease activity. Each of first 5 questions was scored by participant on 100 mm scale, range 0=none to 100=very severe, higher scores = more severe disease activity. Sixth question: duration of morning stiffness, was on scale for 0=0 hours to 100=2 hours, higher scores = larger duration of morning stiffness. BASDAI score obtained by computing mean score for 2 questions related to morning stiffness (Q5 [severity of morning stiffness], Q6 [duration of morning stiffness]) and adding that value to sum of scores for first 4Q and then dividing total by 5. BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5. BASDAI total score ranged from 0 to 10, higher scores = more severe disease activity. Reported values were converted to cm for analysis. The improvement was relative to period 2 baseline(last visit before treatment withdrawal).
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 28, 32, 40, 48, 56, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 112
  Week 28 | 77.7 [69.33 to 84.62]
  Week 32: number analyzed (Participants) | 94
  Week 32 | 77.7 [68.48 to 85.16]
  Week 40: number analyzed (Participants) | 69
  Week 40 | 73.9 [62.72 to 83.14]
  Week 48: number analyzed (Participants) | 53
  Week 48 | 77.4 [64.84 to 86.98]
  Week 56: number analyzed (Participants) | 42
  Week 56 | 83.3 [70.04 to 92.22]
  Week 64: number analyzed (Participants) | 34
  Week 64 | 76.5 [60.45 to 88.20]

77. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): Observed Cases (OC): Period 3
Description: 50% improvement from baseline in BASDAI: percentage of participants who achieved 50% decrease from baseline in their BASDAI total score. BASDAI consisted: 6 questions (Q) related to disease activity. Each of first 5 questions was scored by participant on 100 mm scale, range 0=none to 100=very severe, higher scores = more severe disease activity. Sixth question: duration of morning stiffness, was on scale for 0=0 hours to 100=2 hours, higher scores = larger duration of morning stiffness. BASDAI score was obtained by computing mean score for 2 questions related to morning stiffness (Q5 [severity of morning stiffness], Q6 [duration of morning stiffness]) and adding that value to sum of the scores for first 4Q and then dividing total by 5. BASDAI=(Q1+Q2+Q3+Q4+(Q5+Q6)/2)/5. BASDAI total score ranged from 0 to 10, higher scores = more severe disease activity. Reported values were converted to cm for analysis. The improvement was relative to period 3 baseline (last visit before retreatment).
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 68, 72, 76
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 20.0 [5.98 to 44.36]
  Week 68: number analyzed (Participants) | 85
  Week 68 | 72.9 [62.84 to 81.51]
  Week 72 | 78.2 [68.65 to 85.83]
  Week 76: number analyzed (Participants) | 85
  Week 76 | 84.7 [75.95 to 91.15]

78. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) :Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 75
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 208
percentage of participants
  Week 4 | 33.7 [27.49 to 40.27]
  Week 8 | 50.5 [43.72 to 57.23]
  Week 12 | 55.8 [48.98 to 62.40]
  Week 16 | 63.9 [57.26 to 70.24]
  Week 24 | 75.0 [68.80 to 80.51]

79. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) :Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 76
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 28, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 28: number analyzed (Participants) | 112
  Week 28 | 77.7 [69.33 to 84.62]
  Week 32 | 67.0 [58.02 to 75.05]
  Week 40 | 57.4 [48.26 to 66.15]
  Week 48 | 51.3 [42.23 to 60.31]
  Week 56 | 47.0 [38.01 to 56.06]
  Week 64 | 41.7 [33.02 to 50.86]

80. Secondary Outcome: Percentage of Participants Who Achieved at Least 50% Improvement From Baseline in Disease Activity According to Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) :Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 77
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 68, 72, 76
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 87
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 20.0 [5.98 to 44.36]
  Week 68: number analyzed (Participants) | 86
  Week 68 | 72.1 [62.00 to 80.73]
  Week 72 | 78.2 [68.65 to 85.83]
  Week 78 | 82.8 [73.82 to 89.56]

81. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Observed Cases (OC): Period 1
Description: Change from baseline in hsCRP levels were reported. hsCRP is a sensitive laboratory assay for serum levels of C-Reactive Protein, which is a biomarker of inflammation.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Etanercept
Number analyzed (Participants) | 209
milligram per liter (mg/L)
  Baseline | 12.73 (20.63)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -8.72 (19.70)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -9.20 (19.68)
  Change at week 12: number analyzed (Participants) | 197
  Change at week 12 | -8.98 (19.92)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -9.12 (20.23)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -9.73 (19.39)

82. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Observed Cases (OC): Period 2
Description: as for outcome 81
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 115
mg/L
  Period 2 Baseline | 1.45 (1.54)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -7.46 (15.23)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 2.60 (5.76)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -6.94 (16.83)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 4.72 (12.31)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 1 Baseline | -5.87 (13.89)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 2 Baseline | 3.04 (6.95)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -5.94 (14.65)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 3.29 (6.83)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -6.31 (12.65)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 2.29 (4.93)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -6.47 (13.43)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 2.38 (5.04)

83. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Observed Cases (OC): Period 3
Description: as for outcome 81
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 87
mg/L
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 7.14 (11.88)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -2.58 (14.89)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 9.15 (21.38)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 1.61 (4.68)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 1 Baseline | -8.20 (16.77)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 2 Baseline | 0.54 (3.11)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 82
  Change at Week 68 from Period 3 Baseline | -4.52 (9.23)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 1 Baseline | -8.21 (16.69)
  Change at Week 72 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 2 Baseline | 0.50 (4.38)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 72 from Period 3 Baseline | -4.46 (9.34)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -7.40 (15.98)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 1.39 (5.65)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 83
  Change at Week 76 from Period 3 Baseline | -3.49 (8.27)

84. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 81
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 209
mg/L
  Baseline | 12.73 (20.63)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -8.72 (19.70)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -9.14 (19.59)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -8.77 (19.66)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -8.72 (19.76)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -9.28 (18.90)

85. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 81
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 115
mg/L
  Period 2 Baseline | 1.45 (1.54)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 1 Baseline | -7.46 (15.23)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 111
  Change at Week 28 from Period 2 Baseline | 2.60 (5.76)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 1 Baseline | -5.86 (15.73)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 32 from Period 2 Baseline | 4.46 (11.24)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 1 Baseline | -5.56 (13.91)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 40 from Period 2 Baseline | 4.76 (10.88)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 1 Baseline | -4.83 (14.26)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 48 from Period 2 Baseline | 5.49 (11.51)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 1 Baseline | -5.05 (14.01)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 56 from Period 2 Baseline | 5.27 (11.13)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 1 Baseline | -4.90 (13.88)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 114
  Change at Week 64 from Period 2 Baseline | 5.42 (11.28)

86. Secondary Outcome: Mean Change From Baseline in Highly Sensitive C Reactive Protein (hsCRP): Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 81
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Etanercept
Number analyzed (Participants) | 87
mg/L
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 7.14 (11.88)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -2.58 (14.89)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 9.15 (21.38)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 3 Baseline | 1.61 (4.68)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -7.98 (16.80)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.53 (9.66)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 83
  Change at Week 68 from Period 3 Baseline | -4.32 (9.34)
  Change at Week 72 from Period 1 Baseline | -7.99 (16.71)
  Change at Week 72 from Period 2 Baseline | 1.47 (10.05)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 72 from Period 3 Baseline | -4.27 (9.45)
  Change at Week 76 from Period 1 Baseline | -7.12 (15.93)
  Change at Week 76 from Period 2 Baseline | 2.34 (10.56)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 3 Baseline | -3.38 (8.36)

87. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 12, 24: Observed Cases (OC): Period 1
Description: The EQ-5D questionnaire is a health-related quality of life assessment (HRQOL). The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a VAS with response options. Overall EQ 5D VAS score ranged from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. In this outcome measure, data for percentage of participants who reached the cut-off value of > 82 is reported. This threshold was based on participant's demographic characteristics and population norm. The outcome measure was planned to be analyzed at baseline, Week 12 and 24.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 209
percentage of participants
  Baseline | 4.3 [2.15 to 7.71]
  Week 12: number analyzed (Participants) | 207
  Week 12 | 28.5 [22.68 to 34.92]
  Week 24: number analyzed (Participants) | 191
  Week 24 | 50.3 [43.21 to 57.30]

88. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: The EQ-5D questionnaire is a HRQOL. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a VAS with response options. Overall EQ 5D VAS score ranged from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. In this outcome measure, data for percentage of participants who reached the cut-off value of > 82 is reported. This threshold was based on participant's demographic characteristics and population norm.
Time Frame: Week 32, 48, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: number analyzed (Participants) | 107
  Week 32 | 43.0 [33.90 to 52.45]
  Week 48: number analyzed (Participants) | 66
  Week 48 | 37.9 [26.90 to 49.90]
  Week 64: number analyzed (Participants) | 41
  Week 64 | 46.3 [31.76 to 61.42]

89. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 88
Time Frame: Week 64, 76
Population: Full analysis set for Period 3 included all participants who took study retreatment medication and had at least one evaluation after restarting active therapy. Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 6.7 [0.73 to 27.18]
  Week 76 | 50.0 [39.58 to 60.42]

90. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: The EQ-5D questionnaire is a HRQOL. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a VAS with response options. Overall EQ 5D VAS score ranged from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. In this outcome measure, data for percentage of participants who reached the cut-off value of > 82 is reported. This threshold was based on participant's demographic characteristics and population norm. This outcome measure was planned to be analyzed at baseline, Week 12 and 24.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 209
percentage of participants
  Baseline | 4.3 [2.15 to 7.71]
  Week 12: number analyzed (Participants) | 207
  Week 12 | 28.5 [22.68 to 34.92]
  Week 24: number analyzed (Participants) | 207
  Week 24 | 47.8 [41.09 to 54.62]

91. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 88
Time Frame: Week 32, 48, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: number analyzed (Participants) | 107
  Week 32 | 43.0 [33.90 to 52.45]
  Week 48: number analyzed (Participants) | 108
  Week 48 | 32.4 [24.14 to 41.61]
  Week 64: number analyzed (Participants) | 108
  Week 64 | 28.7 [20.82 to 37.71]

92. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) VAS Score > 82 at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 88
Time Frame: Week 64, 76
Population: FAS Period 3: all participants who took study retreatment medication and had at least one evaluation after restarting active therapy. Missing data was imputed using mixed LOCF. Overall Number of Participants Analyzed" = participants who were evaluable for this outcome measure and "number analyzed" = participants evaluable at specific time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 6.7 [0.73 to 27.18]
  Week 76 | 50.0 [39.58 to 60.42]

93. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 12, 24: Observed Cases (OC): Period 1
Description: The EuroQol-5D is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=severe problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "no problem" and 0 representing ''worst health condition''. This outcome measure was planned to be analyzed at baseline, Week 12 and 24.
Time Frame: Week 12, 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 207
percentage of participants
  Week 12 | 70.0 [63.56 to 75.98]
  Week 24: number analyzed (Participants) | 191
  Week 24 | 79.1 [72.88 to 84.37]

94. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: The EuroQol-5D is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=severe problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "no problem" and 0 representing ''worst health condition''.
Time Frame: Week 32, 48, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: number analyzed (Participants) | 107
  Week 32 | 72.0 [62.95 to 79.81]
  Week 48: number analyzed (Participants) | 66
  Week 48 | 68.2 [56.35 to 78.46]
  Week 64: number analyzed (Participants) | 41
  Week 64 | 75.6 [61.03 to 86.71]

95. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 94
Time Frame: Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 53.3 [29.39 to 76.12]
  Week 76 | 82.6 [73.53 to 89.44]

96. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 93
Time Frame: Week 12, 24
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 207
percentage of participants
  Week 12 | 70.0 [63.56 to 75.98]
  Week 24 | 76.8 [70.72 to 82.16]

97. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 94
Time Frame: Week 32, 48, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: number analyzed (Participants) | 107
  Week 32 | 72.0 [62.95 to 79.81]
  Week 48: number analyzed (Participants) | 108
  Week 48 | 62.0 [52.66 to 70.77]
  Week 64: number analyzed (Participants) | 108
  Week 64 | 61.1 [51.72 to 69.91]

98. Secondary Outcome: Percentage of Participants With >=0.05 Score Increase From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Score at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 94
Time Frame: Week 64, 76
Population: as for outcome 92
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 53.3 [29.39 to 76.12]
  Week 76 | 82.6 [73.53 to 89.44]

99. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 12, 24: Observed Cases (OC): Period 1
Description: as for outcome 93
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 209
percentage of participants
  Baseline: mobility | 32.5 [26.46 to 39.09]
  Baseline: self-care | 64.6 [57.94 to 70.84]
  Baseline: usual activity | 20.6 [15.52 to 26.44]
  Baseline: pain/discomfort | 1.9 [0.65 to 4.49]
  Baseline: anxiety/depression | 37.3 [30.97 to 44.02]
  Week 12: mobility: number analyzed (Participants) | 207
  Week 12: mobility | 65.2 [58.55 to 71.46]
  Week 12: self-care: number analyzed (Participants) | 207
  Week 12: self-care | 86.5 [81.32 to 90.62]
  Week 12: usual activity: number analyzed (Participants) | 207
  Week 12: usual activity | 48.3 [41.56 to 55.10]
  Week 12: pain/discomfort: number analyzed (Participants) | 207
  Week 12: pain/discomfort | 25.6 [20.03 to 31.86]
  Week 12: anxiety/depression: number analyzed (Participants) | 207
  Week 12: anxiety/depression | 64.7 [58.06 to 71.00]
  Week 24: mobility: number analyzed (Participants) | 191
  Week 24: mobility | 80.6 [74.59 to 85.75]
  Week 24: self-care: number analyzed (Participants) | 191
  Week 24: self-care | 93.2 [88.96 to 96.13]
  Week 24: usual activity: number analyzed (Participants) | 191
  Week 24: usual activity | 64.4 [57.43 to 70.93]
  Week 24: pain/discomfort: number analyzed (Participants) | 191
  Week 24: pain/discomfort | 44.0 [37.07 to 51.06]
  Week 24: anxiety/depression: number analyzed (Participants) | 191
  Week 24: anxiety/depression | 78.0 [71.74 to 83.44]

100. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 94
Time Frame: Week 32, 48, 64
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: mobility: number analyzed (Participants) | 107
  Week 32: mobility | 66.4 [57.06 to 74.78]
  Week 32: self-care: number analyzed (Participants) | 107
  Week 32: self-care | 83.2 [75.25 to 89.34]
  Week 32: usual activity: number analyzed (Participants) | 107
  Week 32: usual activity | 55.1 [45.68 to 64.32]
  Week 32: pain/discomfort: number analyzed (Participants) | 107
  Week 32: pain/discomfort | 28.0 [20.19 to 37.05]
  Week 32: anxiety/depression: number analyzed (Participants) | 107
  Week 32: anxiety/depression | 70.1 [60.97 to 78.15]
  Week 48: mobility: number analyzed (Participants) | 66
  Week 48: mobility | 71.2 [59.56 to 81.05]
  Week 48: self-care: number analyzed (Participants) | 66
  Week 48: self-care | 87.9 [78.43 to 94.10]
  Week 48: usual activity: number analyzed (Participants) | 66
  Week 48: usual activity | 66.7 [54.77 to 77.14]
  Week 48: pain/discomfort: number analyzed (Participants) | 66
  Week 48: pain/discomfort | 31.8 [21.54 to 43.65]
  Week 48: anxiety/depression: number analyzed (Participants) | 66
  Week 48: anxiety/depression | 69.7 [57.95 to 79.76]
  Week 64: mobility: number analyzed (Participants) | 41
  Week 64: mobility | 68.3 [53.18 to 80.92]
  Week 64: self-care: number analyzed (Participants) | 41
  Week 64: self-care | 85.4 [72.30 to 93.65]
  Week 64: usual activity: number analyzed (Participants) | 41
  Week 64: usual activity | 63.4 [48.17 to 76.84]
  Week 64: pain/discomfort: number analyzed (Participants) | 41
  Week 64: pain/discomfort | 34.1 [21.10 to 49.35]
  Week 64: anxiety/depression: number analyzed (Participants) | 41
  Week 64: anxiety/depression | 73.2 [58.37 to 84.83]

101. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 94
Time Frame: Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: mobility: number analyzed (Participants) | 15
  Week 64: mobility | 26.7 [9.74 to 51.66]
  Week 64: self-care: number analyzed (Participants) | 15
  Week 64: self-care | 73.3 [48.34 to 90.26]
  Week 64: usual activity: number analyzed (Participants) | 15
  Week 64: usual activity | 26.7 [9.74 to 51.66]
  Week 64: pain/discomfort: number analyzed (Participants) | 15
  Week 64: pain/discomfort | 6.7 [0.73 to 27.18]
  Week 64: anxiety/depression: number analyzed (Participants) | 15
  Week 64: anxiety/depression | 46.7 [23.88 to 70.61]
  Week 76: mobility | 73.3 [63.24 to 81.73]
  Week 76: self-care | 93.0 [86.19 to 97.04]
  Week 76: usual activity | 61.6 [51.10 to 71.38]
  Week 76: pain/discomfort | 40.7 [30.76 to 51.25]
  Week 76: anxiety/depression | 75.6 [65.76 to 83.71]

102. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 93
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 209
percentage of participants
  Baseline: mobility | 32.5 [26.46 to 39.09]
  Baseline: self-care | 64.6 [57.94 to 70.84]
  Baseline: usual activity | 20.6 [15.52 to 26.44]
  Baseline: pain/discomfort | 1.9 [0.65 to 4.49]
  Baseline: anxiety/depression | 37.3 [30.97 to 44.02]
  Week 12: mobility: number analyzed (Participants) | 207
  Week 12: mobility | 65.2 [58.55 to 71.46]
  Week 12: self-care: number analyzed (Participants) | 207
  Week 12: self-care | 86.5 [81.32 to 90.62]
  Week 12: usual activity: number analyzed (Participants) | 207
  Week 12: usual activity | 48.3 [41.56 to 55.10]
  Week 12: pain/discomfort: number analyzed (Participants) | 207
  Week 12: pain/discomfort | 25.6 [20.03 to 31.86]
  Week 12: anxiety/depression: number analyzed (Participants) | 207
  Week 12: anxiety/depression | 64.7 [58.06 to 71.00]
  Week 24: mobility: number analyzed (Participants) | 207
  Week 24: mobility | 77.3 [71.23 to 82.60]
  Week 24: self-care: number analyzed (Participants) | 207
  Week 24: self-care | 91.8 [87.46 to 94.95]
  Week 24: usual activity: number analyzed (Participants) | 207
  Week 24: usual activity | 61.4 [54.60 to 67.79]
  Week 24: pain/discomfort: number analyzed (Participants) | 207
  Week 24: pain/discomfort | 41.1 [34.52 to 47.85]
  Week 24: anxiety/depression: number analyzed (Participants) | 207
  Week 24: anxiety/depression | 75.8 [69.68 to 81.29]

103. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 94
Time Frame: Week 32, 48, 64
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 115
percentage of participants
  Week 32: mobility: number analyzed (Participants) | 107
  Week 32: mobility | 66.4 [57.06 to 74.78]
  Week 32: self-care: number analyzed (Participants) | 107
  Week 32: self-care | 83.2 [75.25 to 89.34]
  Week 32: usual activity: number analyzed (Participants) | 107
  Week 32: usual activity | 55.1 [45.68 to 64.32]
  Week 32: pain/discomfort: number analyzed (Participants) | 107
  Week 32: pain/discomfort | 28.0 [20.19 to 37.05]
  Week 32: anxiety/depression: number analyzed (Participants) | 107
  Week 32: anxiety/depression | 70.1 [60.97 to 78.15]
  Week 48: mobility: number analyzed (Participants) | 108
  Week 48: mobility | 57.4 [47.99 to 66.44]
  Week 48: self-care: number analyzed (Participants) | 108
  Week 48: self-care | 77.8 [69.27 to 84.82]
  Week 48: usual activity: number analyzed (Participants) | 108
  Week 48: usual activity | 51.9 [42.48 to 61.12]
  Week 48: pain/discomfort: number analyzed (Participants) | 108
  Week 48: pain/discomfort | 22.2 [15.18 to 30.73]
  Week 48: anxiety/depression: number analyzed (Participants) | 108
  Week 48: anxiety/depression | 66.7 [57.43 to 75.03]
  Week 64: mobility: number analyzed (Participants) | 108
  Week 64: mobility | 51.9 [42.48 to 61.12]
  Week 64: self-care: number analyzed (Participants) | 108
  Week 64: self-care | 72.2 [63.27 to 80.00]
  Week 64: usual activity: number analyzed (Participants) | 108
  Week 64: usual activity | 44.4 [35.32 to 53.86]
  Week 64: pain/discomfort: number analyzed (Participants) | 108
  Week 64: pain/discomfort | 16.7 [10.56 to 24.53]
  Week 64: anxiety/depression: number analyzed (Participants) | 108
  Week 64: anxiety/depression | 65.7 [56.47 to 74.18]

104. Secondary Outcome: Percentage of Participants Who Achieved an European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Score of 1 at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 94
Time Frame: Week 64, 76
Population: as for outcome 92
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 86
percentage of participants
  Week 64: mobility: number analyzed (Participants) | 15
  Week 64: mobility | 26.7 [9.74 to 51.66]
  Week 64: self-care: number analyzed (Participants) | 15
  Week 64: self-care | 73.3 [48.34 to 90.26]
  Week 64: usual activity: number analyzed (Participants) | 15
  Week 64: usual activity | 26.7 [9.74 to 51.66]
  Week 64: pain/discomfort: number analyzed (Participants) | 15
  Week 64: pain/discomfort | 6.7 [0.73 to 27.18]
  Week 64: anxiety/depression: number analyzed (Participants) | 15
  Week 64: anxiety/depression | 46.7 [23.88 to 70.61]
  Week 76: mobility | 73.3 [63.24 to 81.73]
  Week 76: self-care | 93.0 [86.19 to 97.04]
  Week 76: usual activity | 61.6 [51.10 to 71.38]
  Week 76: pain/discomfort | 40.7 [30.76 to 51.25]
  Week 76: anxiety/depression | 75.6 [65.76 to 83.71]

105. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 12, 24: Observed Cases (OC): Period 1
Description: as for outcome 94
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 0.42 (0.35)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | 0.30 (0.35)
  Change at week 24: number analyzed (Participants) | 191
  Change at week 24 | 0.38 (0.37)

106. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 94
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.89 (0.14)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | 0.27 (0.35)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | -0.15 (0.24)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 1 Baseline | 0.26 (0.32)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 2 Baseline | -0.13 (0.25)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 1 Baseline | 0.25 (0.28)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 2 Baseline | -0.12 (0.22)

107. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 94
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Period 3 Baseline (last visit before retreatment), Week 64, 76
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 0.55 (0.27)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | 0.17 (0.51)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -0.29 (0.27)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.01 (0.12)
  Change at Week 76 from Period 1 Baseline | 0.43 (0.37)
  Change at Week 76 from Period 2 Baseline | -0.06 (0.15)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | 0.27 (0.31)

108. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 94
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 0.42 (0.35)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | 0.30 (0.35)
  Change at week 24: number analyzed (Participants) | 207
  Change at week 24 | 0.37 (0.37)

109. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 94
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.89 (0.14)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | 0.27 (0.35)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | -0.15 (0.24)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 1 Baseline | 0.24 (0.33)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 2 Baseline | -0.18 (0.27)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 1 Baseline | 0.21 (0.30)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 2 Baseline | -0.21 (0.27)

110. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Index Scores at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 94
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 0.55 (0.27)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | 0.17 (0.51)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -0.29 (0.27)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.01 (0.12)
  Change at Week 76 from Period 1 Baseline | 0.43 (0.37)
  Change at Week 76 from Period 2 Baseline | -0.06 (0.15)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | 0.27 (0.31)

111. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 12, 24: Observed Cases (OC): Period 1
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores (physical component scores [PCS]; mental component scores [MCS]). Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value).
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 193
units on a scale
  Baseline | 33.29 (7.13)
  Change at week 12: number analyzed (Participants) | 185
  Change at week 12 | 8.84 (8.54)
  Change at week 24: number analyzed (Participants) | 173
  Change at week 24 | 12.90 (9.30)

112. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores: PCS, MCS. Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value).
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: Full analysis set for Period 2 included all participants who had at least one evaluation during period 2. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 114
units on a scale
  Period 2 Baseline | 50.03 (6.96)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 96
  Change at Week 32 from Period 1 Baseline | 9.62 (10.50)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 102
  Change at Week 32 from Period 2 Baseline | -5.97 (9.07)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 59
  Change at Week 48 from Period 1 Baseline | 8.02 (9.53)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 64
  Change at Week 48 from Period 2 Baseline | -7.84 (8.72)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 39
  Change at Week 64 from Period 1 Baseline | 9.18 (9.34)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 40
  Change at Week 64 from Period 2 Baseline | -7.17 (9.32)

113. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 112
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 82
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 77
  Period 3 Baseline | 34.39 (7.16)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -0.81 (9.87)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -16.06 (9.61)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | -2.98 (3.72)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 74
  Change at Week 76 from Period 1 Baseline | 11.76 (7.84)
  Change at Week 76 from Period 2 Baseline | -3.21 (5.47)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 73
  Change at Week 76 from Period 3 Baseline | 11.36 (8.61)

114. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 112
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 193
units on a scale
  Baseline | 33.29 (7.13)
  Change at week 12: number analyzed (Participants) | 185
  Change at week 12 | 8.84 (8.54)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | 12.14 (9.37)

115. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 112
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: Full analysis set for Period 2 included all participants who had at least one evaluation during period 2. Missing data was imputed using mixed LOCF. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 114
units on a scale
  Period 2 Baseline | 50.03 (6.96)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 96
  Change at Week 32 from Period 1 Baseline | 9.62 (10.50)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 102
  Change at Week 32 from Period 2 Baseline | -5.97 (9.07)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 99
  Change at Week 48 from Period 1 Baseline | 6.52 (10.40)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 105
  Change at Week 48 from Period 2 Baseline | -9.19 (9.37)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 99
  Change at Week 64 from Period 1 Baseline | 5.52 (10.57)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 105
  Change at Week 64 from Period 2 Baseline | -10.32 (9.64)

116. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 112
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 82
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 77
  Period 3 Baseline | 34.39 (7.16)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -0.81 (9.87)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -16.06 (9.61)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | -2.98 (3.72)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 74
  Change at Week 76 from Period 1 Baseline | 11.76 (7.84)
  Change at Week 76 from Period 2 Baseline | -3.21 (5.47)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 73
  Change at Week 76 from Period 3 Baseline | 11.36 (8.61)

117. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 12, 24: Period 1
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores: PCS, MCS. Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value). The improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 197
percentage of participants
  Week 12 | 73.1 [66.60 to 78.92]
  Week 24: number analyzed (Participants) | 186
  Week 24 | 79.6 [73.35 to 84.88]

118. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 32, 48, 64: Period 2
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores: PCS, MCS. Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value). Improvement was relative to period 2 baseline (last visit before treatment withdrawal).
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 103
percentage of participants
  Week 32 | 72.8 [63.68 to 80.69]
  Week 48: number analyzed (Participants) | 64
  Week 48 | 70.3 [58.41 to 80.42]
  Week 64: number analyzed (Participants) | 40
  Week 64 | 75.0 [60.17 to 86.36]

119. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 64, 76: Period 3
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores: PCS, MCS. Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value). Improvement was relative to period 3 baseline (last visit before retreatment).
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 82
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 26.7 [9.74 to 51.66]
  Week 76 | 80.5 [70.94 to 87.93]

120. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 12, 24: Period 1
Description: as for outcome 117
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 197
percentage of participants
  Week 12 | 62.4 [55.53 to 68.98]
  Week 24: number analyzed (Participants) | 186
  Week 24 | 73.7 [67.00 to 79.59]

121. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 32, 48, 64: Period 2
Description: as for outcome 118
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 103
percentage of participants
  Week 32 | 65.0 [55.53 to 73.74]
  Week 48: number analyzed (Participants) | 64
  Week 48 | 59.4 [47.15 to 70.78]
  Week 64: number analyzed (Participants) | 40
  Week 64 | 62.5 [47.05 to 76.21]

122. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Physical Component Score at Week 64, 76: Period 3
Description: as for outcome 119
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 82
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 20.0 [5.98 to 44.36]
  Week 76 | 74.4 [64.21 to 82.88]

123. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 12, 24: Observed Cases (OC): Period 1
Description: as for outcome 112
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 193
units on a scale
  Baseline | 44.23 (10.69)
  Change at week 12: number analyzed (Participants) | 185
  Change at week 12 | 5.24 (9.36)
  Change at week 24: number analyzed (Participants) | 173
  Change at week 24 | 9.23 (10.52)

124. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 112
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 114
units on a scale
  Period 2 Baseline | 55.06 (6.33)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 96
  Change at Week 32 from Period 1 Baseline | 5.71 (10.19)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 102
  Change at Week 32 from Period 2 Baseline | -3.74 (8.00)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 59
  Change at Week 48 from Period 1 Baseline | 6.36 (9.36)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 64
  Change at Week 48 from Period 2 Baseline | -3.19 (7.68)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 39
  Change at Week 64 from Period 1 Baseline | 4.99 (9.14)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 40
  Change at Week 64 from Period 2 Baseline | -3.86 (8.39)

125. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 112
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 82
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 77
  Period 3 Baseline | 47.95 (9.16)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | 0.92 (8.80)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -7.66 (9.63)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.46 (4.25)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 74
  Change at Week 76 from Period 1 Baseline | 8.81 (9.87)
  Change at Week 76 from Period 2 Baseline | -2.13 (7.00)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 73
  Change at Week 76 from Period 3 Baseline | 4.24 (7.61)

126. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 112
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 193
units on a scale
  Baseline | 44.23 (10.69)
  Change at week 12: number analyzed (Participants) | 185
  Change at week 12 | 5.24 (9.36)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | 8.39 (10.69)

127. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 112
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 115
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 114
units on a scale
  Period 2 Baseline | 55.06 (6.33)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 96
  Change at Week 32 from Period 1 Baseline | 5.71 (10.19)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 102
  Change at Week 32 from Period 2 Baseline | -3.74 (8.00)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 99
  Change at Week 48 from Period 1 Baseline | 5.83 (9.15)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 105
  Change at Week 48 from Period 2 Baseline | -3.99 (8.14)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 99
  Change at Week 64 from Period 1 Baseline | 5.17 (9.15)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 105
  Change at Week 64 from Period 2 Baseline | -4.84 (8.31)

128. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 112
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 82
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 77
  Period 3 Baseline | 47.95 (9.16)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | 0.92 (8.80)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | -7.66 (9.63)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.46 (4.25)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 74
  Change at Week 76 from Period 1 Baseline | 8.81 (9.87)
  Change at Week 76 from Period 2 Baseline | -2.13 (7.00)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 73
  Change at Week 76 from Period 3 Baseline | 4.24 (7.61)

129. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 12, 24: Period 1
Description: SF-36 is widely used generic quality of life instrument that assesses the participant's general health and functional status. SF-36 consists of 36 questions that grouped into 8 domains (physical functioning, vitality, social functioning, mental health, role physical, bodily pain, role emotional and general health). Domain scores range from 0 (worst value) to 100 (best value), with greater scores reflecting better health status. Scores of 8 health aspects were summarized to derive the 2 component scores: PCS, MCS. Four domains of the SF-36 comprises the PCS score (physical functioning, role-physical, bodily pain, and general health) and remaining 4 domains comprises of the MCS score (vitality, social functioning, role-emotional, and mental health). Each PCS and MCS are scored from 0 to 100 with higher scores indicating better health (0= worst value and 100= best value). Improvement was relative to baseline (Day 1).
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 197
percentage of participants
  Week 12 | 52.8 [45.82 to 59.68]
  Week 24: number analyzed (Participants) | 186
  Week 24 | 67.2 [60.23 to 73.65]

130. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 32, 48, 64: Period 2
Description: as for outcome 118
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 103
percentage of participants
  Week 32 | 59.2 [49.59 to 68.35]
  Week 48: number analyzed (Participants) | 64
  Week 48 | 54.7 [42.51 to 66.45]
  Week 64: number analyzed (Participants) | 40
  Week 64 | 60.0 [44.56 to 74.05]

131. Secondary Outcome: Percentage of Participants With >=2.5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 64, 76: Period 3
Description: as for outcome 119
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 82
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 26.7 [9.74 to 51.66]
  Week 76 | 64.6 [53.92 to 74.33]

132. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 12, 24: Period 1
Description: as for outcome 117
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 197
percentage of participants
  Week 12 | 45.2 [38.34 to 52.16]
  Week 24: number analyzed (Participants) | 186
  Week 24 | 59.7 [52.52 to 66.53]

133. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 32, 48, 64: Period 2
Description: as for outcome 118
Time Frame: Period 2 baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 103
percentage of participants
  Week 32 | 48.5 [39.04 to 58.12]
  Week 48: number analyzed (Participants) | 64
  Week 48 | 45.3 [33.55 to 57.49]
  Week 64: number analyzed (Participants) | 40
  Week 64 | 40.0 [25.95 to 55.44]

134. Secondary Outcome: Percentage of Participants With >=5 Score Improvement From Baseline in Short Form-36 (SF-36) Mental Component Score (MCS) at Week 64, 76: Period 3
Description: as for outcome 119
Time Frame: Period 3 baseline (last visit before retreatment), Week 64, 76
Population: as for outcome 89
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 82
percentage of participants
  Week 64: number analyzed (Participants) | 15
  Week 64 | 6.7 [0.73 to 27.18]
  Week 76 | 56.1 [45.30 to 66.47]

135. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Observed Cases (OC): Period 1
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem here "ankylosing spondylitis (AS)" affected work attendance, work productivity and productivity in non-work regular activities. Participants were asked to consider the past 7 days prior to each questionnaire day. The questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, and percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: FAS for Period 1 included all participants who took study medication and had one evaluation after baseline. Here, "Overall Number of Participants Analyzed" included participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 140
units on a scale
  Baseline | 50.79 (28.13)
  Change at week 4: number analyzed (Participants) | 133
  Change at week 4 | -15.19 (23.82)
  Change at week 8: number analyzed (Participants) | 125
  Change at week 8 | -21.44 (27.58)
  Change at week 12: number analyzed (Participants) | 115
  Change at week 12 | -21.83 (30.13)
  Change at week 16: number analyzed (Participants) | 120
  Change at week 16 | -27.58 (27.62)
  Change at week 24: number analyzed (Participants) | 118
  Change at week 24 | -35.08 (27.14)

136. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Observed Cases (OC): Period 2
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which a specified health problem here "AS" affected work attendance, work productivity and productivity in non-work regular activities. Participants were asked to consider the past 7 days prior to each questionnaire day. The questionnaire asks: current employment status, hours worked, hours missed from work for any reason other than AS, hours missed from work due to AS, degree to which AS affected work productivity, and degree to a which AS affected non-work regular activities. Four component scores were then calculated: percent work time missed due to AS; percent impairment while working due to AS, percent overall work impairment due to AS, and percent non-work activity impairment due to AS. The computed percentage range for each sub-scale was from 0-100, with higher numbers indicating greater impairment and less productivity.
Time Frame: as for outcome 28
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 92
units on a scale
  Period 2 Baseline | 10.11 (13.05)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 77
  Change at Week 28 from Period 1 Baseline | -31.56 (32.37)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 83
  Change at Week 28 from Period 2 Baseline | 6.87 (18.67)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 60
  Change at Week 32 from Period 1 Baseline | -31.00 (30.35)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 32 from Period 2 Baseline | 9.70 (19.21)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 49
  Change at Week 40 from Period 1 Baseline | -25.71 (32.40)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 51
  Change at Week 40 from Period 2 Baseline | 14.12 (24.99)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 35
  Change at Week 48 from Period 1 Baseline | -22.86 (31.58)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 36
  Change at Week 48 from Period 2 Baseline | 20.56 (26.07)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 28
  Change at Week 56 from Period 1 Baseline | -32.14 (30.11)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 31
  Change at Week 56 from Period 2 Baseline | 6.77 (21.35)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 24
  Change at Week 64 from Period 1 Baseline | -19.17 (26.53)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 26
  Change at Week 64 from Period 2 Baseline | 20.77 (37.19)

137. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Observed Cases (OC): Period 3
Description: as for outcome 136
Time Frame: as for outcome 32
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 67
units on a scale
  Period 3 Baseline | 45.37 (29.20)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 10
  Change at Week 64 from Period 1 Baseline | 8.00 (33.93)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 2 Baseline | 43.64 (22.48)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 10
  Change at Week 64 from Period 3 Baseline | 13.00 (30.57)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 57
  Change at Week 68 from Period 1 Baseline | -26.32 (30.86)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 60
  Change at Week 68 from Period 2 Baseline | 13.67 (22.09)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 60
  Change at Week 68 from Period 3 Baseline | -22.83 (25.78)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 59
  Change at Week 72 from Period 1 Baseline | -32.03 (29.58)
  Change at Week 72 from Period 2 Baseline: number analyzed (Participants) | 64
  Change at Week 72 from Period 2 Baseline | 7.97 (18.10)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 63
  Change at Week 72 from Period 3 Baseline | -29.05 (23.88)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 59
  Change at Week 76 from Period 1 Baseline | -34.41 (27.68)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 62
  Change at Week 76 from Period 2 Baseline | 6.45 (13.92)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 61
  Change at Week 76 from Period 3 Baseline | -30.49 (26.55)

138. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 136
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: FAS for Period 1 included all participants who took study medication and had one evaluation after baseline. Missing data was imputed using mixed LOCF .Here, "Overall Number of Participants Analyzed" included participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 140
units on a scale
  Baseline | 50.79 (28.13)
  Change at week 4: number analyzed (Participants) | 133
  Change at week 4 | -15.19 (23.82)
  Change at week 8: number analyzed (Participants) | 136
  Change at week 8 | -21.25 (27.36)
  Change at week 12: number analyzed (Participants) | 137
  Change at week 12 | -20.44 (29.18)
  Change at week 16: number analyzed (Participants) | 137
  Change at week 16 | -24.53 (28.31)
  Change at week 24: number analyzed (Participants) | 137
  Change at week 24 | -29.93 (29.27)

139. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 136
Time Frame: as for outcome 28
Population: as for outcome 115
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 92
units on a scale
  Period 2 Baseline | 10.11 (13.05)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 77
  Change at Week 28 from Period 1 Baseline | -31.56 (32.37)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 83
  Change at Week 28 from Period 2 Baseline | 6.87 (18.67)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 79
  Change at Week 32 from Period 1 Baseline | -24.94 (34.34)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 32 from Period 2 Baseline | 13.41 (21.36)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 79
  Change at Week 40 from Period 1 Baseline | -19.87 (35.68)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 40 from Period 2 Baseline | 18.12 (24.76)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 79
  Change at Week 48 from Period 1 Baseline | -17.22 (35.26)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 48 from Period 2 Baseline | 20.71 (25.49)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 79
  Change at Week 56 from Period 1 Baseline | -17.97 (35.13)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 87
  Change at Week 56 from Period 2 Baseline | 19.43 (25.76)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 79
  Change at Week 64 from Period 1 Baseline | -12.91 (33.97)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 87
  Change at Week 64 from Period 2 Baseline | 25.06 (29.49)

140. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 136
Time Frame: as for outcome 32
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 67
units on a scale
  Period 3 Baseline | 45.37 (29.20)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 10
  Change at Week 64 from Period 1 Baseline | 8.00 (33.93)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 2 Baseline | 43.64 (22.48)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 10
  Change at Week 64 from Period 3 Baseline | 13.00 (30.57)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 59
  Change at Week 68 from Period 1 Baseline | -25.25 (30.98)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 63
  Change at Week 68 from Period 2 Baseline | 14.92 (22.35)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 63
  Change at Week 68 from Period 3 Baseline | -22.06 (25.41)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 60
  Change at Week 72 from Period 1 Baseline | -31.67 (29.47)
  Change at Week 72 from Period 2 Baseline: number analyzed (Participants) | 65
  Change at Week 72 from Period 2 Baseline | 8.46 (18.39)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 64
  Change at Week 72 from Period 3 Baseline | -28.44 (24.18)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 60
  Change at Week 76 from Period 1 Baseline | -33.83 (27.81)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 65
  Change at Week 76 from Period 2 Baseline | 6.46 (13.74)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 64
  Change at Week 76 from Period 3 Baseline | -29.69 (26.24)

141. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 24: Last Observation Carried Forward (LOCF): Period 1
Description: Change from baseline in MRI score of spine was assessed using SPARCC method. Scoring was based on 6 consecutive coronal slices from posterior to anterior. Each joint was divided into 4 quadrants. Each quadrant was assigned score of 0=no lesion or 1=increased signal. This part of coring allows for total score ranging from 0-8 for the 2 joints of one coronal slice. For each slice, score was increased by 1 for each joint that exhibits an intense signal in any quadrant (thereby allowing for an increase of up to 2 points in total score for each slice). Also, for each slice, an additional score of 1 was given for each joint that includes a lesion demonstrating continuous increased signal of depth >=1 cm from articular surface (thereby allowing for an additional increase of up to 2 points for each slice). The total minimum and maximum score for all joints across 6 slices was 0 to 72 where higher scores reflecting worse disease.
Time Frame: Baseline (Day 1 Week 1), Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 204
units on a scale
  Baseline | 8.48 (12.83)
  Change at week 24: number analyzed (Participants) | 143
  Change at week 24 | -6.08 (11.71)

142. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 141
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 48, 64
Population: as for outcome 115
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 68
units on a scale
  Period 2 Baseline | 2.41 (3.59)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -6.04 (12.99)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 29
  Change at Week 48 from Period 2 Baseline | 2.07 (5.32)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 37
  Change at Week 64 from Period 1 Baseline | -6.81 (13.74)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 29
  Change at Week 64 from Period 2 Baseline | 1.45 (4.43)

143. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 141
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 78
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 50
  Period 3 Baseline | 3.98 (7.28)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -5.17 (8.16)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 4
  Change at Week 64 from Period 2 Baseline | -2.00 (3.37)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 4
  Change at Week 64 from Period 3 Baseline | 4.75 (11.53)
  Change at Week 76 from Period 1 Baseline | -8.44 (12.92)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 44
  Change at Week 76 from Period 2 Baseline | -1.41 (3.28)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 46
  Change at Week 76 from Period 3 Baseline | -1.96 (8.84)

144. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 24: Observed Cases (OC): Period 1
Description: as for outcome 141
Time Frame: Baseline (Day 1 Week 1), Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 204
units on a scale
  Baseline | 8.48 (12.83)
  Change at week 24: number analyzed (Participants) | 143
  Change at week 24 | -6.08 (11.71)

145. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 141
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 48, 64
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 68
units on a scale
  Period 2 Baseline | 2.41 (3.59)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -6.04 (12.99)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 29
  Change at Week 48 from Period 2 Baseline | 2.07 (5.32)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 27
  Change at Week 64 from Period 1 Baseline | -5.96 (13.83)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 19
  Change at Week 64 from Period 2 Baseline | 0.37 (1.12)

146. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score) at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 141
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 78
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 50
  Period 3 Baseline | 3.98 (7.28)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -5.17 (8.16)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 4
  Change at Week 64 from Period 2 Baseline | -2.00 (3.37)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 4
  Change at Week 64 from Period 3 Baseline | 4.75 (11.53)
  Change at Week 76 from Period 1 Baseline | -8.44 (12.92)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 44
  Change at Week 76 from Period 2 Baseline | -1.41 (3.28)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 46
  Change at Week 76 from Period 3 Baseline | -1.96 (8.84)

147. Secondary Outcome: Time to Ankylosing Spondylitis Disease Activity Score (ASDAS) Inactive Disease After Re-treatment in Period 3
Description: Time to ASDAS inactive disease was defined as the time from first dose of retreatment until the first observed event of ASDAS inactive disease. Inactive disease is defined as an ASDAS score <1.3. for ASDAS-CRP or ASDAS score of >=2.1 for ASDAS-ESR. Participants who did not achieve ASDAS inactive disease were censored at the time of the last ASDAS evaluation in the interval.
Time Frame: Within 12 weeks of Period 3 (retreatment period from Week 64 to 76)
Population: Full analysis set for Period 3 included all participants who took study retreatment medication and had at least one evaluation after restarting active therapy.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Etanercept
Number analyzed (Participants) | 87
weeks | 5.1 [4.29 to 8.14]

148. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 1
Description: Participants assessed their overall disease activity over the last 48 hours by using a 100 mm pain scale that ranges from 0 mm (none) to 100 mm (severe pain), where higher scores indicated more pain. The reported values then converted to cm for analysis purposes.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 6.34 (2.14)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.48 (2.45)
  Change at week 8: number analyzed (Participants) | 201
  Change at week 8 | -3.06 (2.71)
  Change at week 12: number analyzed (Participants) | 198
  Change at week 12 | -3.44 (2.74)
  Change at week 16: number analyzed (Participants) | 192
  Change at week 16 | -3.90 (2.74)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -4.72 (2.71)

149. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 2
Description: as for outcome 148
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.61 (0.57)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -4.08 (3.01)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 1.46 (2.47)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 1 Baseline | -3.87 (3.07)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 94
  Change at Week 32 from Period 2 Baseline | 1.68 (2.49)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 1 Baseline | -3.62 (2.90)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 2 Baseline | 1.74 (2.47)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -3.65 (2.73)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 1.81 (2.70)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -3.67 (2.63)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 1.48 (2.45)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -3.07 (3.01)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.66 (2.95)

150. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 3
Description: as for outcome 148
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline | 6.27 (2.24)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.26 (4.09)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.95 (2.35)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 0.67 (2.48)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -4.21 (2.64)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.63 (1.90)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 3 Baseline | -4.09 (2.63)
  Change at Week 72 from Period 1 Baseline | -4.60 (2.59)
  Change at Week 72 from Period 2 Baseline | 1.23 (1.87)
  Change at Week 72 from Period 3 Baseline | -4.44 (2.64)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -4.91 (2.50)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 1.01 (1.42)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 3 Baseline | -4.75 (2.49)

151. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 148
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 6.34 (2.14)
  Change at week 4: number analyzed (Participants) | 208
  Change at week 4 | -2.48 (2.45)
  Change at week 8: number analyzed (Participants) | 208
  Change at week 8 | -3.04 (2.69)
  Change at week 12: number analyzed (Participants) | 208
  Change at week 12 | -3.35 (2.74)
  Change at week 16: number analyzed (Participants) | 208
  Change at week 16 | -3.70 (2.80)
  Change at week 24: number analyzed (Participants) | 208
  Change at week 24 | -4.45 (2.87)

152. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 148
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.61 (0.57)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 1 Baseline | -4.08 (3.01)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 112
  Change at Week 28 from Period 2 Baseline | 1.46 (2.47)
  Change at Week 32 from Period 1 Baseline | -3.24 (3.33)
  Change at Week 32 from Period 2 Baseline | 2.27 (2.81)
  Change at Week 40 from Period 1 Baseline | -2.73 (3.29)
  Change at Week 40 from Period 2 Baseline | 2.79 (2.92)
  Change at Week 48 from Period 1 Baseline | -2.33 (3.22)
  Change at Week 48 from Period 2 Baseline | 3.18 (2.99)
  Change at Week 56 from Period 1 Baseline | -2.09 (3.13)
  Change at Week 56 from Period 2 Baseline | 3.42 (3.00)
  Change at Week 64 from Period 1 Baseline | -1.81 (3.10)
  Change at Week 64 from Period 2 Baseline | 3.71 (3.04)

153. Secondary Outcome: Change From Baseline in Subject Assessment of Disease Activity (SADA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 148
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline | 6.27 (2.24)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.26 (4.09)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.95 (2.35)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 3 Baseline | 0.67 (2.48)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 1 Baseline | -4.17 (2.66)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.66 (1.91)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 3 Baseline | -4.03 (2.66)
  Change at Week 72 from Period 1 Baseline | -4.60 (2.59)
  Change at Week 72 from Period 2 Baseline | 1.23 (1.87)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 3 Baseline | -4.44 (2.64)
  Change at Week 76 from Period 1 Baseline | -4.83 (2.54)
  Change at Week 76 from Period 2 Baseline | 1.01 (1.43)
  Change at Week 76 from Period 3 Baseline | -4.66 (2.52)

154. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 1
Description: The physician assessed the overall disease activity of participants over the last 48 hours by using a 100 mm VAS pain scale that ranges from 0 mm (none) to 100 mm (severe pain), where higher scores indicated more pain. The reported values then converted to cm for analysis purposes.
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 208
cm
  Baseline | 6.07 (1.88)
  Change at week 4: number analyzed (Participants) | 207
  Change at week 4 | -2.89 (2.41)
  Change at week 8: number analyzed (Participants) | 200
  Change at week 8 | -3.83 (2.52)
  Change at week 12: number analyzed (Participants) | 196
  Change at week 12 | -4.16 (2.41)
  Change at week 16: number analyzed (Participants) | 191
  Change at week 16 | -4.57 (2.39)
  Change at week 24: number analyzed (Participants) | 189
  Change at week 24 | -4.81 (2.26)

155. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 2
Description: as for outcome 154
Time Frame: as for outcome 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.63 (0.82)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 109
  Change at Week 28 from Period 1 Baseline | -4.65 (2.50)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 2 Baseline | 0.92 (1.69)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 1 Baseline | -4.27 (2.61)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 93
  Change at Week 32 from Period 2 Baseline | 1.33 (1.92)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 1 Baseline | -3.98 (3.22)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 69
  Change at Week 40 from Period 2 Baseline | 1.59 (2.07)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 1 Baseline | -4.78 (2.45)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 53
  Change at Week 48 from Period 2 Baseline | 1.24 (1.97)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 1 Baseline | -4.67 (2.45)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 56 from Period 2 Baseline | 1.16 (1.79)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 1 Baseline | -4.22 (2.63)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 34
  Change at Week 64 from Period 2 Baseline | 1.40 (2.42)

156. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Observed Cases (OC): Period 3
Description: as for outcome 154
Time Frame: as for outcome 32
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 4.89 (1.99)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -2.18 (2.91)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.52 (1.85)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 13
  Change at Week 64 from Period 3 Baseline | 1.88 (2.21)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 1 Baseline | -4.51 (2.15)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 2 Baseline | 1.06 (1.31)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 83
  Change at Week 68 from Period 3 Baseline | -3.17 (2.09)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 1 Baseline | -4.89 (1.92)
  Change at Week 72 from Period 2 Baseline | 0.70 (1.09)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 72 from Period 3 Baseline | -3.52 (2.25)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 1 Baseline | -5.25 (1.98)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 2 Baseline | 0.34 (0.83)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 83
  Change at Week 76 from Period 3 Baseline | -3.95 (2.22)

157. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 154
Time Frame: Baseline (Day 1 Week 1), Week 4, 8, 12, 16, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 208
cm
  Baseline | 6.07 (1.88)
  Change at week 4: number analyzed (Participants) | 207
  Change at week 4 | -2.89 (2.41)
  Change at week 8: number analyzed (Participants) | 207
  Change at week 8 | -3.76 (2.61)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | -4.02 (2.56)
  Change at week 16: number analyzed (Participants) | 207
  Change at week 16 | -4.32 (2.58)
  Change at week 24: number analyzed (Participants) | 207
  Change at week 24 | -4.54 (2.51)

158. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 154
Time Frame: as for outcome 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 0.63 (0.82)
  Change at Week 28 from Period 1 Baseline: number analyzed (Participants) | 109
  Change at Week 28 from Period 1 Baseline | -4.65 (2.50)
  Change at Week 28 from Period 2 Baseline: number analyzed (Participants) | 110
  Change at Week 28 from Period 2 Baseline | 0.92 (1.69)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 32 from Period 1 Baseline | -3.91 (2.69)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 32 from Period 2 Baseline | 1.64 (2.11)
  Change at Week 40 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 40 from Period 1 Baseline | -3.31 (3.04)
  Change at Week 40 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 40 from Period 2 Baseline | 2.24 (2.31)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 48 from Period 1 Baseline | -3.15 (3.00)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 48 from Period 2 Baseline | 2.40 (2.43)
  Change at Week 56 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 56 from Period 1 Baseline | -2.89 (2.93)
  Change at Week 56 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 56 from Period 2 Baseline | 2.65 (2.40)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 112
  Change at Week 64 from Period 1 Baseline | -2.66 (2.88)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 113
  Change at Week 64 from Period 2 Baseline | 2.88 (2.53)

159. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) Visual Analogue Scale (VAS): Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 154
Time Frame: as for outcome 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 87
cm
  Period 3 Baseline: number analyzed (Participants) | 85
  Period 3 Baseline | 4.89 (1.99)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 14
  Change at Week 64 from Period 1 Baseline | -2.18 (2.91)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 4.52 (1.85)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 13
  Change at Week 64 from Period 3 Baseline | 1.88 (2.21)
  Change at Week 68 from Period 1 Baseline: number analyzed (Participants) | 85
  Change at Week 68 from Period 1 Baseline | -4.46 (2.19)
  Change at Week 68 from Period 2 Baseline: number analyzed (Participants) | 86
  Change at Week 68 from Period 2 Baseline | 1.12 (1.42)
  Change at Week 68 from Period 3 Baseline: number analyzed (Participants) | 84
  Change at Week 68 from Period 3 Baseline | -3.10 (2.18)
  Change at Week 72 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 72 from Period 1 Baseline | -4.89 (1.92)
  Change at Week 72 from Period 2 Baseline | 0.70 (1.09)
  Change at Week 72 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 72 from Period 3 Baseline | -3.52 (2.25)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 86
  Change at Week 76 from Period 1 Baseline | -5.22 (1.99)
  Change at Week 76 from Period 2 Baseline | 0.37 (0.89)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 85
  Change at Week 76 from Period 3 Baseline | -3.85 (2.27)

160. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: The BAS-G was a 2-question assessment evaluating the effect of AS on the participants well-being over the last week and last 6 months. Each question scored by the participant on a 100 mm VAS scale ranging from 0 (very Good) to 100 (very Bad), where higher scores indicated worse health condition. The total BAS-G score calculated as the average scores of these two questions and then converted into cm for analysis. Total BAS-G score ranged from 0 to 10 cm, where higher scores indicated worse health condition.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 6.48 (1.93)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | -2.58 (2.25)
  Change at week 24: number analyzed (Participants) | 207
  Change at week 24 | -3.95 (2.64)

161. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score) at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 160
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 1.39 (1.49)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | -3.78 (2.79)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | 1.10 (2.22)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 1 Baseline | -3.04 (2.80)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 2 Baseline | 1.84 (2.46)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 1 Baseline | -2.64 (2.72)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 2 Baseline | 2.24 (2.58)

162. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 160
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 86
cm
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 4.74 (2.02)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -2.23 (2.41)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 2.94 (1.81)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.83 (2.16)
  Change at Week 76 from Period 1 Baseline | -4.35 (2.46)
  Change at Week 76 from Period 2 Baseline | 0.57 (1.74)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | -2.53 (2.10)

163. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score at Week 12, 24: Observed Cases (OC): Period 1
Description: as for outcome 160
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 209
cm
  Baseline | 6.48 (1.93)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | -2.58 (2.25)
  Change at week 24: number analyzed (Participants) | 191
  Change at week 24 | -4.11 (2.62)

164. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score) at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 160
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 115
cm
  Period 2 Baseline | 1.39 (1.49)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | -3.78 (2.79)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | 1.10 (2.22)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 1 Baseline | -3.54 (2.51)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 2 Baseline | 1.44 (2.37)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 1 Baseline | -3.52 (2.51)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 2 Baseline | 1.58 (2.55)

165. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Global Index (BAS-G) Score at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 160
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Etanercept
Number analyzed (Participants) | 86
cm
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 4.74 (2.02)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -2.23 (2.41)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 2.94 (1.81)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.83 (2.16)
  Change at Week 76 from Period 1 Baseline | -4.35 (2.46)
  Change at Week 76 from Period 2 Baseline | 0.57 (1.74)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | -2.53 (2.10)

166. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 12, 24: Observed Cases (OC): Period 1
Description: Number of swollen joints was determined by examination of 44 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling =0, swelling =1.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 147
swollen joints
  Baseline | 2.32 (3.01)
  Change at week 12: number analyzed (Participants) | 91
  Change at week 12 | -1.72 (3.36)
  Change at week 24: number analyzed (Participants) | 60
  Change at week 24 | -1.85 (3.82)

167. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 166
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 77
swollen joints
  Period 2 Baseline | 0.95 (1.89)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 1 Baseline | -2.69 (3.28)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 2 Baseline | 0.46 (1.79)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 22
  Change at Week 48 from Period 1 Baseline | -1.64 (2.40)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 22
  Change at Week 48 from Period 2 Baseline | -0.59 (2.20)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 1 Baseline | -0.82 (2.27)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 2 Baseline | 0.36 (2.62)

168. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 166
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 42
swollen joints
  Period 3: baseline | 1.19 (1.76)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -0.67 (1.03)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 2 Baseline | 1.17 (2.48)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 3
  Change at Week 64 from Period 3 Baseline | 0.33 (1.53)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 1 Baseline | -2.50 (3.13)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 2 Baseline | 0.50 (1.34)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 17
  Change at Week 76 from Period 3 Baseline | -0.88 (1.96)

169. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 166
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 147
swollen joints
  Baseline | 2.32 (3.01)
  Change at week 12: number analyzed (Participants) | 91
  Change at week 12 | -1.72 (3.36)
  Change at week 24: number analyzed (Participants) | 96
  Change at week 24 | -1.92 (3.52)

170. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 166
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 115
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 77
swollen joints
  Period 2 Baseline | 0.95 (1.89)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 1 Baseline | -2.69 (3.28)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 2 Baseline | 0.46 (1.79)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 48 from Period 1 Baseline | -2.24 (3.00)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 48 from Period 2 Baseline | -0.02 (2.17)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 47
  Change at Week 64 from Period 1 Baseline | -2.00 (3.05)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 47
  Change at Week 64 from Period 2 Baseline | 0.04 (2.37)

171. Secondary Outcome: Change From Baseline in Number of Swollen Joint Count at Week 64, 76 : Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 166
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Etanercept
Number analyzed (Participants) | 42
swollen joints
  Period 3 Baseline | 1.19 (1.76)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -0.67 (1.03)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 2 Baseline | 1.17 (2.48)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 3
  Change at Week 64 from Period 3 Baseline | 0.33 (1.53)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 19
  Change at Week 76 from Period 1 Baseline | -2.32 (3.15)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 19
  Change at Week 76 from Period 2 Baseline | 0.53 (1.31)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 3 Baseline | -0.72 (2.02)

172. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 12, 24: Observed Cases (OC): Period 1
Description: Number of tender joints was determined by examining 44 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 147
tender joints
  Baseline | 5.96 (5.44)
  Change at week 12: number analyzed (Participants) | 91
  Change at week 12 | -2.82 (4.86)
  Change at week 24: number analyzed (Participants) | 60
  Change at week 24 | -3.67 (5.72)

173. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 172
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 77
tender joints
  Period 2 Baseline | 2.70 (2.58)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 1 Baseline | -3.27 (4.65)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 2 Baseline | 0.61 (2.70)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 22
  Change at Week 48 from Period 1 Baseline | -2.68 (3.71)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 22
  Change at Week 48 from Period 2 Baseline | -0.73 (3.56)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 1 Baseline | -2.27 (2.28)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 11
  Change at Week 64 from Period 2 Baseline | 0.18 (3.74)

174. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 64, 76: : Observed Cases (OC): Period 3
Description: as for outcome 172
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 42
tender joints
  Period 3 Baseline | 3.60 (2.80)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -0.17 (1.47)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 2 Baseline | 0.33 (1.97)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 3
  Change at Week 64 from Period 3 Baseline | 0.00 (2.00)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 1 Baseline | -3.56 (2.91)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 2 Baseline | 0.06 (1.63)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 17
  Change at Week 76 from Period 3 Baseline | -1.94 (2.41)

175. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 172
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 147
tender joints
  Baseline | 5.96 (5.44)
  Change at week 12: number analyzed (Participants) | 91
  Change at week 12 | -2.82 (4.86)
  Change at week 24: number analyzed (Participants) | 96
  Change at week 24 | -3.15 (5.26)

176. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 172
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 115
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 77
tender joints
  Period 2 Baseline | 2.70 (2.58)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 1 Baseline | -3.27 (4.65)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 26
  Change at Week 32 from Period 2 Baseline | 0.61 (2.70)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 48 from Period 1 Baseline | -2.88 (4.11)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 48 from Period 2 Baseline | -0.05 (3.37)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 47
  Change at Week 64 from Period 1 Baseline | -2.72 (3.81)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 47
  Change at Week 64 from Period 2 Baseline | -0.09 (3.47)

177. Secondary Outcome: Change From Baseline in Number of Tender Joint Count at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 172
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Etanercept
Number analyzed (Participants) | 42
tender joints
  Period 3 Baseline | 3.60 (2.80)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 1 Baseline | -0.17 (1.47)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 6
  Change at Week 64 from Period 2 Baseline | 0.33 (1.97)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 3
  Change at Week 64 from Period 3 Baseline | 0.00 (2.00)
  Change at Week 76 from Period 1 Baseline: number analyzed (Participants) | 19
  Change at Week 76 from Period 1 Baseline | -3.32 (3.02)
  Change at Week 76 from Period 2 Baseline: number analyzed (Participants) | 19
  Change at Week 76 from Period 2 Baseline | 0.11 (1.59)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 18
  Change at Week 76 from Period 3 Baseline | -1.72 (2.52)

178. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 12, 24: Observed Cases (OC): Period 1
Description: Dactylitis is the inflammation of finger and/or toe joints (digits). Dactylitis scores was calculated by evaluating each of the 10 fingers and 10 toes. Each digit was evaluated on a 4-point scale ranging from of 0 to 3 where 0 = none, 1= mild, 2 = moderate, 3 = severe inflammation. The total score was calculated as the sum of scores for the 20 digits, total score ranged from 0 to 60, where higher scores indicated severe inflammation.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 0.42 (1.43)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | -0.27 (1.45)
  Change at week 24: number analyzed (Participants) | 191
  Change at week 24 | -0.30 (1.44)

179. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 178
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.02 (0.13)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | -0.42 (1.32)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | 0.01 (0.22)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 1 Baseline | -0.36 (1.26)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 2 Baseline | 0.09 (0.74)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 42
  Change at Week 64 from Period 1 Baseline | -0.57 (1.61)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 42
  Change at Week 64 from Period 2 Baseline | 0.07 (0.34)

180. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 178
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 0.08 (0.35)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.33 (1.05)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 0.20 (0.56)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.25 (0.71)
  Change at Week 76 from Period 1 Baseline | -0.50 (1.47)
  Change at Week 76 from Period 2 Baseline | 0.00 (0.15)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | -0.06 (0.37)

181. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 178
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 209
units on a scale
  Baseline | 0.42 (1.43)
  Change at week 12: number analyzed (Participants) | 207
  Change at week 12 | -0.27 (1.45)
  Change at week 24: number analyzed (Participants) | 207
  Change at week 24 | -0.28 (1.38)

182. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 178
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.02 (0.13)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 1 Baseline | -0.42 (1.32)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 32 from Period 2 Baseline | 0.01 (0.22)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 1 Baseline | -0.36 (1.24)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 48 from Period 2 Baseline | 0.06 (0.62)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 1 Baseline | -0.39 (1.28)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 108
  Change at Week 64 from Period 2 Baseline | 0.04 (0.30)

183. Secondary Outcome: Change From Baseline in Dactylitis Total Score at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 178
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 80
  Period 3 Baseline | 0.08 (0.35)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -0.33 (1.05)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 0.20 (0.56)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 8
  Change at Week 64 from Period 3 Baseline | 0.25 (0.71)
  Change at Week 76 from Period 1 Baseline | -0.50 (1.47)
  Change at Week 76 from Period 2 Baseline | 0.00 (0.15)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 80
  Change at Week 76 from Period 3 Baseline | -0.06 (0.37)

184. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 12, 24: Observed Cases (OC) : Period 1
Description: The MASES is an index used to measure the severity of enthesitis. Enthesitis is the inflammation of enthuses (heels). The MASES assesses 13 sites for enthesitis. Each site is scored as 0 or 1 depending on whether enthesitis is present or absent. Sites assessed include 1st costochondral joint (left/right), 7 th costochondral joint (l/r), posterior superior iliac spine (l/r), posterior anterior iliac spine (l/r), iliac crest (l/r), proximal insertion of Achilles tendon (l/r) and 5th lumbar spinous process. The MASES is the sum of all site scores range from 0 (no inflammation) to 13 (worst possible inflammation) where higher scores indicate more severe inflammation of entheses.
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 208
units on a scale
  Baseline | 2.86 (2.98)
  Change at week 12: number analyzed (Participants) | 205
  Change at week 12 | -1.22 (2.55)
  Change at week 24: number analyzed (Participants) | 190
  Change at week 24 | -1.59 (2.59)

185. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 32, 48, 64: Observed Cases (OC): Period 2
Description: as for outcome 184
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2 Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.36 (0.97)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 106
  Change at Week 32 from Period 1 Baseline | -1.06 (2.49)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 106
  Change at Week 32 from Period 2 Baseline | 0.71 (1.76)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 1 Baseline | -1.50 (2.48)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 66
  Change at Week 48 from Period 2 Baseline | 0.32 (1.15)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 1 Baseline | -1.37 (2.30)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 41
  Change at Week 64 from Period 2 Baseline | 0.49 (1.00)

186. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 64, 76: Observed Cases (OC): Period 3
Description: as for outcome 184
Time Frame: as for outcome 107
Population: as for outcome 89
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 79
  Period 3 Baseline | 1.48 (1.80)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -1.13 (2.03)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 0.67 (2.13)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 7
  Change at Week 64 from Period 3 Baseline | 0.14 (0.90)
  Change at Week 76 from Period 1 Baseline | -1.86 (2.14)
  Change at Week 76 from Period 2 Baseline | -0.06 (1.13)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 79
  Change at Week 76 from Period 3 Baseline | -1.08 (1.61)

187. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 12, 24: Last Observation Carried Forward (LOCF): Period 1
Description: as for outcome 184
Time Frame: Baseline (Day 1 Week 1), Week 12, 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 208
units on a scale
  Baseline | 2.86 (2.98)
  Change at week 12: number analyzed (Participants) | 205
  Change at week 12 | -1.22 (2.55)
  Change at week 24: number analyzed (Participants) | 206
  Change at week 24 | -1.55 (2.64)

188. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 32, 48, 64: Last Observation Carried Forward (LOCF): Period 2
Description: as for outcome 184
Time Frame: Period 1 Baseline (Day 1 Week 1), Period 2: Baseline (last visit before treatment withdrawal), Week 32, 48, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 115
units on a scale
  Period 2 Baseline | 0.36 (0.97)
  Change at Week 32 from Period 1 Baseline: number analyzed (Participants) | 106
  Change at Week 32 from Period 1 Baseline | -1.06 (2.49)
  Change at Week 32 from Period 2 Baseline: number analyzed (Participants) | 106
  Change at Week 32 from Period 2 Baseline | 0.71 (1.76)
  Change at Week 48 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 48 from Period 1 Baseline | -1.13 (2.47)
  Change at Week 48 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 48 from Period 2 Baseline | 0.62 (1.55)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 107
  Change at Week 64 from Period 1 Baseline | -1.00 (2.24)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 107
  Change at Week 64 from Period 2 Baseline | 0.75 (1.55)

189. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) at Week 64, 76: Last Observation Carried Forward (LOCF): Period 3
Description: as for outcome 184
Time Frame: as for outcome 107
Population: as for outcome 92
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 86
units on a scale
  Period 3 Baseline: number analyzed (Participants) | 79
  Period 3 Baseline | 1.48 (1.80)
  Change at Week 64 from Period 1 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 1 Baseline | -1.13 (2.03)
  Change at Week 64 from Period 2 Baseline: number analyzed (Participants) | 15
  Change at Week 64 from Period 2 Baseline | 0.67 (2.13)
  Change at Week 64 from Period 3 Baseline: number analyzed (Participants) | 7
  Change at Week 64 from Period 3 Baseline | 0.14 (0.90)
  Change at Week 76 from Period 1 Baseline | -1.86 (2.14)
  Change at Week 76 from Period 2 Baseline | -0.06 (1.13)
  Change at Week 76 from Period 3 Baseline: number analyzed (Participants) | 79
  Change at Week 76 from Period 3 Baseline | -1.08 (1.61)

190. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of investigational product and up to 28 days after the last dose of investigational product that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (for period 1: maximum up to 28 weeks, for period 2: maximum up to 68 weeks, period 3: maximum up to 80 weeks)
Population: Safety analysis set for each period included all participants who entered the period and for periods 1 and 3; all participants who received 1 dose of investigational drug.
Measure: Count of Participants; unit: Participants
Groups:
- Etanercept: Period 1: All enrolled participants with nr-ax SpA were treated for 24 weeks with 50 milligram weekly dose of Etanercept in Period 1 (Induction Period). Participants who did not qualify for Period 2 were followed up until 28 days after last dose of Etanercept.
- Etanercept: Period 2: Participants who achieved ASDAS CRP level less than 1.3 at Week 24 then entered into Period 2 (Withdrawal Period). In this period, participants discontinued Etanercept for 40 weeks (from Week 24 to Week 64). Participants who did not qualify for Period 2 were followed up until 28 days after last dose of Etanercept.
- Etanercept: Period 3: Participants who achieved an ASDAS ESR level >= 2.1 by Week 64, then entered into Period 3 (Retreatment Period) of 12 weeks, treated with 50 mg weekly doses, and then followed up until 28 days after last dose of Etanercept.
Arm/Group | Etanercept: Period 1 | Etanercept: Period 2 | Etanercept: Period 3
Number analyzed (Participants) | 209 | 119 | 87
Participants
  AEs | 147 | 37 | 29
  SAEs | 6 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (for period 1: maximum up to 28 weeks, for period 2: maximum up to 68 weeks, period 3: maximum up to 80 weeks)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Etanercept: Period 1 | Etanercept: Period 2 | Etanercept: Period 3
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/119 | 0/87
Serious Adverse Events (participants affected / at risk) | 6/209 | 1/119 | 0/87
Other Adverse Events (participants affected / at risk) | 72/209 | 0/119 | 8/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Period 1 (N=209) | Etanercept: Period 2 (N=119) | Etanercept: Period 3 (N=87)
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Period 1 (N=209) | Etanercept: Period 2 (N=119) | Etanercept: Period 3 (N=87)
Injection site erythema (General disorders) | 15 | 0 | 0
Injection site reaction (General disorders) | 15 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 33 | 0 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT02509026/SAP_000.pdf
  • Study Protocol (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT02509026/Prot_001.pdf